CLINICAL TRIAL: NCT01076959
Title: Humira 40 mg/0.8 mL for Subcutaneous Injection - Drug Use Investigation (All Patient Investigation) for Rheumatoid Arthritis
Brief Title: Drug Use Investigation for Humira® - All Patient Investigation for Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: P10-559
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Results first posted 2012-08-07 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Humira: The sponsor was required to include all patients diagnosed with rheumatoid arthritis and who were treated Humira in routine medical practice during the review period by the PMDA. The safety analysis set included all patients who met all eligibility criteria and received at least one dose of Humira. The full analysis set included all patients who were treated with Humira for at least 2 weeks and had complete DAS 28 assessments at baseline and at least one other time point.

SUMMARY:
To clarify the following matters:

* Unknown adverse reactions (especially clinically significant adverse reactions)
* Incidence and conditions of occurrence of adverse reactions in the clinical setting
* Factors that may affect the safety and effectiveness of Humira

ELIGIBILITY:
Inclusion Criteria:

* All patients prescribed and treated with Humira are included in this survey.

Exclusion Criteria:

* Contraindications according to the Package Insert:

  * Patients who have serious infections,
  * Patients who have tuberculosis,
  * Patients with a history of hypersensitivity to any ingredient of Humira,
  * Patients who have demyelinating disease or with a history of demyelinating disease,
  * Patients who have cardiac failure congestive.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients prescribed and treated with Humira included in this survey.
Sampling Method: Non-Probability Sample
Enrollment: 7972 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toshiro Maeda, Study Director — Abbott Japan Co.,Ltd
Locations (1723):
- Japan (1723):
  - Site Reference ID/Investigator# 35904, Aichi
  - Site Reference ID/Investigator# 35905, Aichi
  - Site Reference ID/Investigator# 35906, Aichi
  - Site Reference ID/Investigator# 35907, Aichi
  - Site Reference ID/Investigator# 35908, Aichi
  - Site Reference ID/Investigator# 35909, Aichi
  - Site Reference ID/Investigator# 35912, Aichi
  - Site Reference ID/Investigator# 35913, Aichi
  - Site Reference ID/Investigator# 35914, Aichi
  - Site Reference ID/Investigator# 35915, Aichi
  - Site Reference ID/Investigator# 35916, Aichi
  - Site Reference ID/Investigator# 35917, Aichi
  - Site Reference ID/Investigator# 35918, Aichi
  - Site Reference ID/Investigator# 35919, Aichi
  - Site Reference ID/Investigator# 35920, Aichi
  - Site Reference ID/Investigator# 35921, Aichi
  - Site Reference ID/Investigator# 35922, Aichi
  - Site Reference ID/Investigator# 35923, Aichi
  - Site Reference ID/Investigator# 35924, Aichi
  - Site Reference ID/Investigator# 36611, Aichi
  - Site Reference ID/Investigator# 36644, Aichi
  - Site Reference ID/Investigator# 36650, Aichi
  - Site Reference ID/Investigator# 36652, Aichi
  - Site Reference ID/Investigator# 36676, Aichi
  - Site Reference ID/Investigator# 36681, Aichi
  - Site Reference ID/Investigator# 36689, Aichi
  - Site Reference ID/Investigator# 36696, Aichi
  - Site Reference ID/Investigator# 36733, Aichi
  - Site Reference ID/Investigator# 36752, Aichi
  - Site Reference ID/Investigator# 36819, Aichi
  - Site Reference ID/Investigator# 36843, Aichi
  - Site Reference ID/Investigator# 36867, Aichi
  - Site Reference ID/Investigator# 36923, Aichi
  - Site Reference ID/Investigator# 36943, Aichi
  - Site Reference ID/Investigator# 36944, Aichi
  - Site Reference ID/Investigator# 36945, Aichi
  - Site Reference ID/Investigator# 39128, Aichi
  - Site Reference ID/Investigator# 39129, Aichi
  - Site Reference ID/Investigator# 39130, Aichi
  - Site Reference ID/Investigator# 39131, Aichi
  - Site Reference ID/Investigator# 39132, Aichi
  - Site Reference ID/Investigator# 39133, Aichi
  - Site Reference ID/Investigator# 39134, Aichi
  - Site Reference ID/Investigator# 39135, Aichi
  - Site Reference ID/Investigator# 39136, Aichi
  - Site Reference ID/Investigator# 39137, Aichi
  - Site Reference ID/Investigator# 39138, Aichi
  - Site Reference ID/Investigator# 39140, Aichi
  - Site Reference ID/Investigator# 39141, Aichi
  - Site Reference ID/Investigator# 39142, Aichi
  - Site Reference ID/Investigator# 39143, Aichi
  - Site Reference ID/Investigator# 39144, Aichi
  - Site Reference ID/Investigator# 39145, Aichi
  - Site Reference ID/Investigator# 39146, Aichi
  - Site Reference ID/Investigator# 39147, Aichi
  - Site Reference ID/Investigator# 39148, Aichi
  - Site Reference ID/Investigator# 39149, Aichi
  - Site Reference ID/Investigator# 39150, Aichi
  - Site Reference ID/Investigator# 39151, Aichi
  - Site Reference ID/Investigator# 39152, Aichi
  - Site Reference ID/Investigator# 39153, Aichi
  - Site Reference ID/Investigator# 39154, Aichi
  - Site Reference ID/Investigator# 39155, Aichi
  - Site Reference ID/Investigator# 39156, Aichi
  - Site Reference ID/Investigator# 39157, Aichi
  - Site Reference ID/Investigator# 39158, Aichi
  - Site Reference ID/Investigator# 39159, Aichi
  - Site Reference ID/Investigator# 39160, Aichi
  - Site Reference ID/Investigator# 39161, Aichi
  - Site Reference ID/Investigator# 39162, Aichi
  - Site Reference ID/Investigator# 39163, Aichi
  - Site Reference ID/Investigator# 39165, Aichi
  - Site Reference ID/Investigator# 39166, Aichi
  - Site Reference ID/Investigator# 39167, Aichi
  - Site Reference ID/Investigator# 39168, Aichi
  - Site Reference ID/Investigator# 42712, Aichi
  - Site Reference ID/Investigator# 42715, Aichi
  - Site Reference ID/Investigator# 42723, Aichi
  - Site Reference ID/Investigator# 42738, Aichi
  - Site Reference ID/Investigator# 42756, Aichi
  - Site Reference ID/Investigator# 42757, Aichi
  - Site Reference ID/Investigator# 42758, Aichi
  - Site Reference ID/Investigator# 42759, Aichi
  - Site Reference ID/Investigator# 42760, Aichi
  - Site Reference ID/Investigator# 42844, Aichi
  - Site Reference ID/Investigator# 42845, Aichi
  - Site Reference ID/Investigator# 42846, Aichi
  - Site Reference ID/Investigator# 42851, Aichi
  - Site Reference ID/Investigator# 42852, Aichi
  - Site Reference ID/Investigator# 58587, Aichi
  - Site Reference ID/Investigator# 58612, Aichi
  - Site Reference ID/Investigator# 58680, Aichi
  - Site Reference ID/Investigator# 58681, Aichi
  - Site Reference ID/Investigator# 58682, Aichi
  - Site Reference ID/Investigator# 58687, Aichi
  - Site Reference ID/Investigator# 58838, Aichi
  - Site Reference ID/Investigator# 58839, Aichi
  - Site Reference ID/Investigator# 58843, Aichi
  - Site Reference ID/Investigator# 58844, Aichi
  - Site Reference ID/Investigator# 58845, Aichi
  - Site Reference ID/Investigator# 58872, Aichi
  - Site Reference ID/Investigator# 39508, Aki Takada
  - Site Reference ID/Investigator# 36549, Akita
  - Site Reference ID/Investigator# 36796, Akita
  - Site Reference ID/Investigator# 36948, Akita
  - Site Reference ID/Investigator# 39169, Akita
  - Site Reference ID/Investigator# 39170, Akita
  - Site Reference ID/Investigator# 39171, Akita
  - Site Reference ID/Investigator# 39172, Akita
  - Site Reference ID/Investigator# 39173, Akita
  - Site Reference ID/Investigator# 42717, Akita
  - Site Reference ID/Investigator# 42871, Akita
  - Site Reference ID/Investigator# 42872, Akita
  - Site Reference ID/Investigator# 58820, Akita
  - Site Reference ID/Investigator# 39865, Amagasaki
  - Site Reference ID/Investigator# 39866, Amagasaki
  - Site Reference ID/Investigator# 35925, Aomori
  - Site Reference ID/Investigator# 35926, Aomori
  - Site Reference ID/Investigator# 35927, Aomori
  - Site Reference ID/Investigator# 39176, Aomori
  - Site Reference ID/Investigator# 39177, Aomori
  - Site Reference ID/Investigator# 39181, Aomori
  - Site Reference ID/Investigator# 39182, Aomori
  - Site Reference ID/Investigator# 39192, Aomori
  - Site Reference ID/Investigator# 42866, Aomori
  - Site Reference ID/Investigator# 42867, Aomori
  - Site Reference ID/Investigator# 42868, Aomori
  - Site Reference ID/Investigator# 58647, Aomori
  - Site Reference ID/Investigator# 58819, Aomori
  - Site Reference ID/Investigator# 36605, Ashiya
  - Site Reference ID/Investigator# 36082, Chiba
  - Site Reference ID/Investigator# 36083, Chiba
  - Site Reference ID/Investigator# 36084, Chiba
  - Site Reference ID/Investigator# 36085, Chiba
  - Site Reference ID/Investigator# 36086, Chiba
  - Site Reference ID/Investigator# 36087, Chiba
  - Site Reference ID/Investigator# 36088, Chiba
  - Site Reference ID/Investigator# 36089, Chiba
  - Site Reference ID/Investigator# 36090, Chiba
  - Site Reference ID/Investigator# 36091, Chiba
  - Site Reference ID/Investigator# 36449, Chiba
  - Site Reference ID/Investigator# 36455, Chiba
  - Site Reference ID/Investigator# 36600, Chiba
  - Site Reference ID/Investigator# 36610, Chiba
  - Site Reference ID/Investigator# 36693, Chiba
  - Site Reference ID/Investigator# 36694, Chiba
  - Site Reference ID/Investigator# 36808, Chiba
  - Site Reference ID/Investigator# 36817, Chiba
  - Site Reference ID/Investigator# 36830, Chiba
  - Site Reference ID/Investigator# 38528, Chiba
  - Site Reference ID/Investigator# 39193, Chiba
  - Site Reference ID/Investigator# 39194, Chiba
  - Site Reference ID/Investigator# 39195, Chiba
  - Site Reference ID/Investigator# 39196, Chiba
  - Site Reference ID/Investigator# 39197, Chiba
  - Site Reference ID/Investigator# 39198, Chiba
  - Site Reference ID/Investigator# 39199, Chiba
  - Site Reference ID/Investigator# 39200, Chiba
  - Site Reference ID/Investigator# 39209, Chiba
  - Site Reference ID/Investigator# 39210, Chiba
  - Site Reference ID/Investigator# 39211, Chiba
  - Site Reference ID/Investigator# 39212, Chiba
  - Site Reference ID/Investigator# 39213, Chiba
  - Site Reference ID/Investigator# 39214, Chiba
  - Site Reference ID/Investigator# 39215, Chiba
  - Site Reference ID/Investigator# 39216, Chiba
  - Site Reference ID/Investigator# 39217, Chiba
  - Site Reference ID/Investigator# 39221, Chiba
  - Site Reference ID/Investigator# 39224, Chiba
  - Site Reference ID/Investigator# 39225, Chiba
  - Site Reference ID/Investigator# 39226, Chiba
  - Site Reference ID/Investigator# 39227, Chiba
  - Site Reference ID/Investigator# 39228, Chiba
  - Site Reference ID/Investigator# 42761, Chiba
  - Site Reference ID/Investigator# 42828, Chiba
  - Site Reference ID/Investigator# 42830, Chiba
  - Site Reference ID/Investigator# 42831, Chiba
  - Site Reference ID/Investigator# 42832, Chiba
  - Site Reference ID/Investigator# 42833, Chiba
  - Site Reference ID/Investigator# 58668, Chiba
  - Site Reference ID/Investigator# 58676, Chiba
  - Site Reference ID/Investigator# 58831, Chiba
  - Site Reference ID/Investigator# 39964, Chūō
  - Site Reference ID/Investigator# 39965, Chūō
  - Site Reference ID/Investigator# 42725, Daisuke
  - Site Reference ID/Investigator# 36092, Ehime
  - Site Reference ID/Investigator# 36093, Ehime
  - Site Reference ID/Investigator# 36903, Ehime
  - Site Reference ID/Investigator# 39229, Ehime
  - Site Reference ID/Investigator# 39230, Ehime
  - Site Reference ID/Investigator# 39231, Ehime
  - Site Reference ID/Investigator# 39234, Ehime
  - Site Reference ID/Investigator# 39235, Ehime
  - Site Reference ID/Investigator# 39239, Ehime
  - Site Reference ID/Investigator# 39240, Ehime
  - Site Reference ID/Investigator# 39241, Ehime
  - Site Reference ID/Investigator# 42740, Ehime
  - Site Reference ID/Investigator# 42815, Ehime
  - Site Reference ID/Investigator# 58592, Ehime
  - Site Reference ID/Investigator# 58601, Ehime
  - Site Reference ID/Investigator# 58778, Ehime
  - Site Reference ID/Investigator# 58779, Ehime
  - Site Reference ID/Investigator# 39910, Fuchū
  - Site Reference ID/Investigator# 42825, Fujisawa
  - Site Reference ID/Investigator# 36094, Fukui
  - Site Reference ID/Investigator# 36095, Fukui
  - Site Reference ID/Investigator# 36096, Fukui
  - Site Reference ID/Investigator# 36097, Fukui
  - Site Reference ID/Investigator# 36548, Fukui
  - Site Reference ID/Investigator# 36571, Fukui
  - Site Reference ID/Investigator# 36742, Fukui
  - Site Reference ID/Investigator# 36911, Fukui
  - Site Reference ID/Investigator# 39246, Fukui
  - Site Reference ID/Investigator# 39247, Fukui
  - Site Reference ID/Investigator# 39248, Fukui
  - Site Reference ID/Investigator# 39252, Fukui
  - Site Reference ID/Investigator# 39253, Fukui
  - Site Reference ID/Investigator# 39254, Fukui
  - Site Reference ID/Investigator# 39255, Fukui
  - Site Reference ID/Investigator# 39256, Fukui
  - Site Reference ID/Investigator# 42762, Fukui
  - Site Reference ID/Investigator# 42924, Fukui
  - Site Reference ID/Investigator# 58595, Fukui
  - Site Reference ID/Investigator# 58611, Fukui
  - Site Reference ID/Investigator# 58706, Fukui
  - Site Reference ID/Investigator# 36099, Fukuoka
  - Site Reference ID/Investigator# 36100, Fukuoka
  - Site Reference ID/Investigator# 36101, Fukuoka
  - Site Reference ID/Investigator# 36102, Fukuoka
  - Site Reference ID/Investigator# 36103, Fukuoka
  - Site Reference ID/Investigator# 36104, Fukuoka
  - Site Reference ID/Investigator# 36105, Fukuoka
  - Site Reference ID/Investigator# 36106, Fukuoka
  - Site Reference ID/Investigator# 36107, Fukuoka
  - Site Reference ID/Investigator# 36108, Fukuoka
  - Site Reference ID/Investigator# 36109, Fukuoka
  - Site Reference ID/Investigator# 36110, Fukuoka
  - Site Reference ID/Investigator# 36111, Fukuoka
  - Site Reference ID/Investigator# 36112, Fukuoka
  - Site Reference ID/Investigator# 36113, Fukuoka
  - Site Reference ID/Investigator# 36114, Fukuoka
  - Site Reference ID/Investigator# 36115, Fukuoka
  - Site Reference ID/Investigator# 36116, Fukuoka
  - Site Reference ID/Investigator# 36118, Fukuoka
  - Site Reference ID/Investigator# 36120, Fukuoka
  - Site Reference ID/Investigator# 36121, Fukuoka
  - Site Reference ID/Investigator# 36122, Fukuoka
  - Site Reference ID/Investigator# 36445, Fukuoka
  - Site Reference ID/Investigator# 36544, Fukuoka
  - Site Reference ID/Investigator# 36568, Fukuoka
  - Site Reference ID/Investigator# 36597, Fukuoka
  - Site Reference ID/Investigator# 36601, Fukuoka
  - Site Reference ID/Investigator# 36606, Fukuoka
  - Site Reference ID/Investigator# 36642, Fukuoka
  - Site Reference ID/Investigator# 36645, Fukuoka
  - Site Reference ID/Investigator# 36651, Fukuoka
  - Site Reference ID/Investigator# 36660, Fukuoka
  - Site Reference ID/Investigator# 36670, Fukuoka
  - Site Reference ID/Investigator# 36692, Fukuoka
  - Site Reference ID/Investigator# 36699, Fukuoka
  - Site Reference ID/Investigator# 36748, Fukuoka
  - Site Reference ID/Investigator# 36799, Fukuoka
  - Site Reference ID/Investigator# 36801, Fukuoka
  - Site Reference ID/Investigator# 36870, Fukuoka
  - Site Reference ID/Investigator# 36907, Fukuoka
  - Site Reference ID/Investigator# 36910, Fukuoka
  - Site Reference ID/Investigator# 36914, Fukuoka
  - Site Reference ID/Investigator# 39174, Fukuoka
  - Site Reference ID/Investigator# 39175, Fukuoka
  - Site Reference ID/Investigator# 39178, Fukuoka
  - Site Reference ID/Investigator# 39179, Fukuoka
  - Site Reference ID/Investigator# 39183, Fukuoka
  - Site Reference ID/Investigator# 39184, Fukuoka
  - Site Reference ID/Investigator# 39185, Fukuoka
  - Site Reference ID/Investigator# 39186, Fukuoka
  - Site Reference ID/Investigator# 39187, Fukuoka
  - Site Reference ID/Investigator# 39188, Fukuoka
  - Site Reference ID/Investigator# 39189, Fukuoka
  - Site Reference ID/Investigator# 39190, Fukuoka
  - Site Reference ID/Investigator# 39191, Fukuoka
  - Site Reference ID/Investigator# 39201, Fukuoka
  - Site Reference ID/Investigator# 39202, Fukuoka
  - Site Reference ID/Investigator# 39203, Fukuoka
  - Site Reference ID/Investigator# 39204, Fukuoka
  - Site Reference ID/Investigator# 39205, Fukuoka
  - Site Reference ID/Investigator# 39206, Fukuoka
  - Site Reference ID/Investigator# 39207, Fukuoka
  - Site Reference ID/Investigator# 39208, Fukuoka
  - Site Reference ID/Investigator# 39218, Fukuoka
  - Site Reference ID/Investigator# 39219, Fukuoka
  - Site Reference ID/Investigator# 39220, Fukuoka
  - Site Reference ID/Investigator# 39222, Fukuoka
  - Site Reference ID/Investigator# 39232, Fukuoka
  - Site Reference ID/Investigator# 39233, Fukuoka
  - Site Reference ID/Investigator# 42711, Fukuoka
  - Site Reference ID/Investigator# 42763, Fukuoka
  - Site Reference ID/Investigator# 42764, Fukuoka
  - Site Reference ID/Investigator# 42805, Fukuoka
  - Site Reference ID/Investigator# 58580, Fukuoka
  - Site Reference ID/Investigator# 58782, Fukuoka
  - Site Reference ID/Investigator# 58786, Fukuoka
  - Site Reference ID/Investigator# 58867, Fukuoka
  - Site Reference ID/Investigator# 58868, Fukuoka
  - Site Reference ID/Investigator# 36002, Fukushima
  - Site Reference ID/Investigator# 36447, Fukushima
  - Site Reference ID/Investigator# 36490, Fukushima
  - Site Reference ID/Investigator# 36649, Fukushima
  - Site Reference ID/Investigator# 36724, Fukushima
  - Site Reference ID/Investigator# 36791, Fukushima
  - Site Reference ID/Investigator# 36821, Fukushima
  - Site Reference ID/Investigator# 36823, Fukushima
  - Site Reference ID/Investigator# 38525, Fukushima
  - Site Reference ID/Investigator# 39236, Fukushima
  - Site Reference ID/Investigator# 39237, Fukushima
  - Site Reference ID/Investigator# 39238, Fukushima
  - Site Reference ID/Investigator# 39242, Fukushima
  - Site Reference ID/Investigator# 39243, Fukushima
  - Site Reference ID/Investigator# 39244, Fukushima
  - Site Reference ID/Investigator# 39245, Fukushima
  - Site Reference ID/Investigator# 39249, Fukushima
  - Site Reference ID/Investigator# 39250, Fukushima
  - Site Reference ID/Investigator# 42720, Fukushima
  - Site Reference ID/Investigator# 42729, Fukushima
  - Site Reference ID/Investigator# 42944, Fukushima
  - Site Reference ID/Investigator# 42945, Fukushima
  - Site Reference ID/Investigator# 42946, Fukushima
  - Site Reference ID/Investigator# 58651, Fukushima
  - Site Reference ID/Investigator# 58823, Fukushima
  - Site Reference ID/Investigator# 36003, Gifu
  - Site Reference ID/Investigator# 36004, Gifu
  - Site Reference ID/Investigator# 36005, Gifu
  - Site Reference ID/Investigator# 36006, Gifu
  - Site Reference ID/Investigator# 36007, Gifu
  - Site Reference ID/Investigator# 36542, Gifu
  - Site Reference ID/Investigator# 36612, Gifu
  - Site Reference ID/Investigator# 36614, Gifu
  - Site Reference ID/Investigator# 36675, Gifu
  - Site Reference ID/Investigator# 36677, Gifu
  - Site Reference ID/Investigator# 36735, Gifu
  - Site Reference ID/Investigator# 36814, Gifu
  - Site Reference ID/Investigator# 36839, Gifu
  - Site Reference ID/Investigator# 36925, Gifu
  - Site Reference ID/Investigator# 36927, Gifu
  - Site Reference ID/Investigator# 36928, Gifu
  - Site Reference ID/Investigator# 36942, Gifu
  - Site Reference ID/Investigator# 36955, Gifu
  - Site Reference ID/Investigator# 39251, Gifu
  - Site Reference ID/Investigator# 39257, Gifu
  - Site Reference ID/Investigator# 39258, Gifu
  - Site Reference ID/Investigator# 39482, Gifu
  - Site Reference ID/Investigator# 39483, Gifu
  - Site Reference ID/Investigator# 39486, Gifu
  - Site Reference ID/Investigator# 39487, Gifu
  - Site Reference ID/Investigator# 39488, Gifu
  - Site Reference ID/Investigator# 39489, Gifu
  - Site Reference ID/Investigator# 39490, Gifu
  - Site Reference ID/Investigator# 42772, Gifu
  - Site Reference ID/Investigator# 42853, Gifu
  - Site Reference ID/Investigator# 42854, Gifu
  - Site Reference ID/Investigator# 42855, Gifu
  - Site Reference ID/Investigator# 42856, Gifu
  - Site Reference ID/Investigator# 42857, Gifu
  - Site Reference ID/Investigator# 42858, Gifu
  - Site Reference ID/Investigator# 58597, Gifu
  - Site Reference ID/Investigator# 58598, Gifu
  - Site Reference ID/Investigator# 58688, Gifu
  - Site Reference ID/Investigator# 58689, Gifu
  - Site Reference ID/Investigator# 58690, Gifu
  - Site Reference ID/Investigator# 58691, Gifu
  - Site Reference ID/Investigator# 58785, Gifu
  - Site Reference ID/Investigator# 58846, Gifu
  - Site Reference ID/Investigator# 58847, Gifu
  - Site Reference ID/Investigator# 58848, Gifu
  - Site Reference ID/Investigator# 58849, Gifu
  - Site Reference ID/Investigator# 58850, Gifu
  - Site Reference ID/Investigator# 36008, Gunma
  - Site Reference ID/Investigator# 36009, Gunma
  - Site Reference ID/Investigator# 36010, Gunma
  - Site Reference ID/Investigator# 36011, Gunma
  - Site Reference ID/Investigator# 36012, Gunma
  - Site Reference ID/Investigator# 36013, Gunma
  - Site Reference ID/Investigator# 36936, Gunma
  - Site Reference ID/Investigator# 36937, Gunma
  - Site Reference ID/Investigator# 39484, Gunma
  - Site Reference ID/Investigator# 39485, Gunma
  - Site Reference ID/Investigator# 39491, Gunma
  - Site Reference ID/Investigator# 39493, Gunma
  - Site Reference ID/Investigator# 39494, Gunma
  - Site Reference ID/Investigator# 39495, Gunma
  - Site Reference ID/Investigator# 39496, Gunma
  - Site Reference ID/Investigator# 39497, Gunma
  - Site Reference ID/Investigator# 39498, Gunma
  - Site Reference ID/Investigator# 39499, Gunma
  - Site Reference ID/Investigator# 42743, Gunma
  - Site Reference ID/Investigator# 42893, Gunma
  - Site Reference ID/Investigator# 42898, Gunma
  - Site Reference ID/Investigator# 42900, Gunma
  - Site Reference ID/Investigator# 42903, Gunma
  - Site Reference ID/Investigator# 58657, Gunma
  - Site Reference ID/Investigator# 39446, Gyōda
  - Site Reference ID/Investigator# 39948, Hagi
  - Site Reference ID/Investigator# 39540, Himeji
  - Site Reference ID/Investigator# 36014, Hiroshima
  - Site Reference ID/Investigator# 36015, Hiroshima
  - Site Reference ID/Investigator# 36016, Hiroshima
  - Site Reference ID/Investigator# 36017, Hiroshima
  - Site Reference ID/Investigator# 36018, Hiroshima
  - Site Reference ID/Investigator# 36019, Hiroshima
  - Site Reference ID/Investigator# 36023, Hiroshima
  - Site Reference ID/Investigator# 36029, Hiroshima
  - Site Reference ID/Investigator# 36744, Hiroshima
  - Site Reference ID/Investigator# 36750, Hiroshima
  - Site Reference ID/Investigator# 36828, Hiroshima
  - Site Reference ID/Investigator# 36840, Hiroshima
  - Site Reference ID/Investigator# 36841, Hiroshima
  - Site Reference ID/Investigator# 38527, Hiroshima
  - Site Reference ID/Investigator# 39500, Hiroshima
  - Site Reference ID/Investigator# 39501, Hiroshima
  - Site Reference ID/Investigator# 39502, Hiroshima
  - Site Reference ID/Investigator# 39503, Hiroshima
  - Site Reference ID/Investigator# 39504, Hiroshima
  - Site Reference ID/Investigator# 39505, Hiroshima
  - Site Reference ID/Investigator# 39506, Hiroshima
  - Site Reference ID/Investigator# 39507, Hiroshima
  - Site Reference ID/Investigator# 39510, Hiroshima
  - Site Reference ID/Investigator# 39516, Hiroshima
  - Site Reference ID/Investigator# 42733, Hiroshima
  - Site Reference ID/Investigator# 42734, Hiroshima
  - Site Reference ID/Investigator# 42841, Hiroshima
  - Site Reference ID/Investigator# 58607, Hiroshima
  - Site Reference ID/Investigator# 58783, Hiroshima
  - Site Reference ID/Investigator# 58792, Hiroshima
  - Site Reference ID/Investigator# 58861, Hiroshima
  - Site Reference ID/Investigator# 58862, Hiroshima
  - Site Reference ID/Investigator# 36021, Hokkaido
  - Site Reference ID/Investigator# 36022, Hokkaido
  - Site Reference ID/Investigator# 36024, Hokkaido
  - Site Reference ID/Investigator# 36026, Hokkaido
  - Site Reference ID/Investigator# 36027, Hokkaido
  - Site Reference ID/Investigator# 36028, Hokkaido
  - Site Reference ID/Investigator# 36130, Hokkaido
  - Site Reference ID/Investigator# 36454, Hokkaido
  - Site Reference ID/Investigator# 36550, Hokkaido
  - Site Reference ID/Investigator# 36579, Hokkaido
  - Site Reference ID/Investigator# 36659, Hokkaido
  - Site Reference ID/Investigator# 36666, Hokkaido
  - Site Reference ID/Investigator# 36667, Hokkaido
  - Site Reference ID/Investigator# 36673, Hokkaido
  - Site Reference ID/Investigator# 36678, Hokkaido
  - Site Reference ID/Investigator# 36804, Hokkaido
  - Site Reference ID/Investigator# 36813, Hokkaido
  - Site Reference ID/Investigator# 36822, Hokkaido
  - Site Reference ID/Investigator# 36958, Hokkaido
  - Site Reference ID/Investigator# 39317, Hokkaido
  - Site Reference ID/Investigator# 39509, Hokkaido
  - Site Reference ID/Investigator# 39511, Hokkaido
  - Site Reference ID/Investigator# 39512, Hokkaido
  - Site Reference ID/Investigator# 39513, Hokkaido
  - Site Reference ID/Investigator# 39515, Hokkaido
  - Site Reference ID/Investigator# 39517, Hokkaido
  - Site Reference ID/Investigator# 39518, Hokkaido
  - Site Reference ID/Investigator# 39519, Hokkaido
  - Site Reference ID/Investigator# 39520, Hokkaido
  - Site Reference ID/Investigator# 39521, Hokkaido
  - Site Reference ID/Investigator# 39522, Hokkaido
  - Site Reference ID/Investigator# 39523, Hokkaido
  - Site Reference ID/Investigator# 39524, Hokkaido
  - Site Reference ID/Investigator# 39525, Hokkaido
  - Site Reference ID/Investigator# 39527, Hokkaido
  - Site Reference ID/Investigator# 39529, Hokkaido
  - Site Reference ID/Investigator# 39530, Hokkaido
  - Site Reference ID/Investigator# 39531, Hokkaido
  - Site Reference ID/Investigator# 39532, Hokkaido
  - Site Reference ID/Investigator# 39533, Hokkaido
  - Site Reference ID/Investigator# 39534, Hokkaido
  - Site Reference ID/Investigator# 39535, Hokkaido
  - Site Reference ID/Investigator# 39539, Hokkaido
  - Site Reference ID/Investigator# 39542, Hokkaido
  - Site Reference ID/Investigator# 39543, Hokkaido
  - Site Reference ID/Investigator# 42714, Hokkaido
  - Site Reference ID/Investigator# 42754, Hokkaido
  - Site Reference ID/Investigator# 42769, Hokkaido
  - Site Reference ID/Investigator# 42770, Hokkaido
  - Site Reference ID/Investigator# 42771, Hokkaido
  - Site Reference ID/Investigator# 42953, Hokkaido
  - Site Reference ID/Investigator# 42954, Hokkaido
  - Site Reference ID/Investigator# 42955, Hokkaido
  - Site Reference ID/Investigator# 42956, Hokkaido
  - Site Reference ID/Investigator# 42957, Hokkaido
  - Site Reference ID/Investigator# 42958, Hokkaido
  - Site Reference ID/Investigator# 42959, Hokkaido
  - Site Reference ID/Investigator# 42960, Hokkaido
  - Site Reference ID/Investigator# 42961, Hokkaido
  - Site Reference ID/Investigator# 58562, Hokkaido
  - Site Reference ID/Investigator# 58569, Hokkaido
  - Site Reference ID/Investigator# 58570, Hokkaido
  - Site Reference ID/Investigator# 58646, Hokkaido
  - Site Reference ID/Investigator# 58800, Hokkaido
  - Site Reference ID/Investigator# 58818, Hokkaido
  - Site Reference ID/Investigator# 36030, Hyōgo
  - Site Reference ID/Investigator# 36031, Hyōgo
  - Site Reference ID/Investigator# 36032, Hyōgo
  - Site Reference ID/Investigator# 36033, Hyōgo
  - Site Reference ID/Investigator# 36034, Hyōgo
  - Site Reference ID/Investigator# 36035, Hyōgo
  - Site Reference ID/Investigator# 36036, Hyōgo
  - Site Reference ID/Investigator# 36037, Hyōgo
  - Site Reference ID/Investigator# 36038, Hyōgo
  - Site Reference ID/Investigator# 36039, Hyōgo
  - Site Reference ID/Investigator# 36040, Hyōgo
  - Site Reference ID/Investigator# 36041, Hyōgo
  - Site Reference ID/Investigator# 36042, Hyōgo
  - Site Reference ID/Investigator# 36043, Hyōgo
  - Site Reference ID/Investigator# 36044, Hyōgo
  - Site Reference ID/Investigator# 36045, Hyōgo
  - Site Reference ID/Investigator# 36046, Hyōgo
  - Site Reference ID/Investigator# 36047, Hyōgo
  - Site Reference ID/Investigator# 36049, Hyōgo
  - Site Reference ID/Investigator# 36053, Hyōgo
  - Site Reference ID/Investigator# 36055, Hyōgo
  - Site Reference ID/Investigator# 36056, Hyōgo
  - Site Reference ID/Investigator# 36451, Hyōgo
  - Site Reference ID/Investigator# 36546, Hyōgo
  - Site Reference ID/Investigator# 36566, Hyōgo
  - Site Reference ID/Investigator# 36604, Hyōgo
  - Site Reference ID/Investigator# 36608, Hyōgo
  - Site Reference ID/Investigator# 36643, Hyōgo
  - Site Reference ID/Investigator# 36647, Hyōgo
  - Site Reference ID/Investigator# 36655, Hyōgo
  - Site Reference ID/Investigator# 36663, Hyōgo
  - Site Reference ID/Investigator# 36686, Hyōgo
  - Site Reference ID/Investigator# 36906, Hyōgo
  - Site Reference ID/Investigator# 36912, Hyōgo
  - Site Reference ID/Investigator# 36922, Hyōgo
  - Site Reference ID/Investigator# 36929, Hyōgo
  - Site Reference ID/Investigator# 39537, Hyōgo
  - Site Reference ID/Investigator# 39538, Hyōgo
  - Site Reference ID/Investigator# 39541, Hyōgo
  - Site Reference ID/Investigator# 39566, Hyōgo
  - Site Reference ID/Investigator# 39567, Hyōgo
  - Site Reference ID/Investigator# 39568, Hyōgo
  - Site Reference ID/Investigator# 39569, Hyōgo
  - Site Reference ID/Investigator# 39579, Hyōgo
  - Site Reference ID/Investigator# 39580, Hyōgo
  - Site Reference ID/Investigator# 39581, Hyōgo
  - Site Reference ID/Investigator# 39858, Hyōgo
  - Site Reference ID/Investigator# 39859, Hyōgo
  - Site Reference ID/Investigator# 39860, Hyōgo
  - Site Reference ID/Investigator# 39861, Hyōgo
  - Site Reference ID/Investigator# 39862, Hyōgo
  - Site Reference ID/Investigator# 39863, Hyōgo
  - Site Reference ID/Investigator# 39867, Hyōgo
  - Site Reference ID/Investigator# 39868, Hyōgo
  - Site Reference ID/Investigator# 39869, Hyōgo
  - Site Reference ID/Investigator# 39870, Hyōgo
  - Site Reference ID/Investigator# 39871, Hyōgo
  - Site Reference ID/Investigator# 39872, Hyōgo
  - Site Reference ID/Investigator# 39873, Hyōgo
  - Site Reference ID/Investigator# 39874, Hyōgo
  - Site Reference ID/Investigator# 39875, Hyōgo
  - Site Reference ID/Investigator# 42719, Hyōgo
  - Site Reference ID/Investigator# 42744, Hyōgo
  - Site Reference ID/Investigator# 42765, Hyōgo
  - Site Reference ID/Investigator# 42767, Hyōgo
  - Site Reference ID/Investigator# 42947, Hyōgo
  - Site Reference ID/Investigator# 42948, Hyōgo
  - Site Reference ID/Investigator# 42949, Hyōgo
  - Site Reference ID/Investigator# 42950, Hyōgo
  - Site Reference ID/Investigator# 42951, Hyōgo
  - Site Reference ID/Investigator# 42952, Hyōgo
  - Site Reference ID/Investigator# 58561, Hyōgo
  - Site Reference ID/Investigator# 58605, Hyōgo
  - Site Reference ID/Investigator# 58704, Hyōgo
  - Site Reference ID/Investigator# 58705, Hyōgo
  - Site Reference ID/Investigator# 58801, Hyōgo
  - Site Reference ID/Investigator# 58854, Hyōgo
  - Site Reference ID/Investigator# 58855, Hyōgo
  - Site Reference ID/Investigator# 36048, Ibaraki
  - Site Reference ID/Investigator# 36050, Ibaraki
  - Site Reference ID/Investigator# 36051, Ibaraki
  - Site Reference ID/Investigator# 36052, Ibaraki
  - Site Reference ID/Investigator# 36054, Ibaraki
  - Site Reference ID/Investigator# 36448, Ibaraki
  - Site Reference ID/Investigator# 36727, Ibaraki
  - Site Reference ID/Investigator# 36805, Ibaraki
  - Site Reference ID/Investigator# 36862, Ibaraki
  - Site Reference ID/Investigator# 36863, Ibaraki
  - Site Reference ID/Investigator# 36865, Ibaraki
  - Site Reference ID/Investigator# 36868, Ibaraki
  - Site Reference ID/Investigator# 36902, Ibaraki
  - Site Reference ID/Investigator# 36908, Ibaraki
  - Site Reference ID/Investigator# 36909, Ibaraki
  - Site Reference ID/Investigator# 39876, Ibaraki
  - Site Reference ID/Investigator# 39877, Ibaraki
  - Site Reference ID/Investigator# 39878, Ibaraki
  - Site Reference ID/Investigator# 39879, Ibaraki
  - Site Reference ID/Investigator# 39880, Ibaraki
  - Site Reference ID/Investigator# 39881, Ibaraki
  - Site Reference ID/Investigator# 39882, Ibaraki
  - Site Reference ID/Investigator# 39883, Ibaraki
  - Site Reference ID/Investigator# 39884, Ibaraki
  - Site Reference ID/Investigator# 39891, Ibaraki
  - Site Reference ID/Investigator# 42753, Ibaraki
  - Site Reference ID/Investigator# 42766, Ibaraki
  - Site Reference ID/Investigator# 42773, Ibaraki
  - Site Reference ID/Investigator# 58652, Ibaraki
  - Site Reference ID/Investigator# 58653, Ibaraki
  - Site Reference ID/Investigator# 58654, Ibaraki
  - Site Reference ID/Investigator# 58824, Ibaraki
  - Site Reference ID/Investigator# 58825, Ibaraki
  - Site Reference ID/Investigator# 42896, Inashiki
  - Site Reference ID/Investigator# 36057, Ishikawa
  - Site Reference ID/Investigator# 36058, Ishikawa
  - Site Reference ID/Investigator# 36061, Ishikawa
  - Site Reference ID/Investigator# 36452, Ishikawa
  - Site Reference ID/Investigator# 36543, Ishikawa
  - Site Reference ID/Investigator# 36918, Ishikawa
  - Site Reference ID/Investigator# 38526, Ishikawa
  - Site Reference ID/Investigator# 39648, Ishikawa
  - Site Reference ID/Investigator# 39651, Ishikawa
  - Site Reference ID/Investigator# 39653, Ishikawa
  - Site Reference ID/Investigator# 39655, Ishikawa
  - Site Reference ID/Investigator# 39888, Ishikawa
  - Site Reference ID/Investigator# 39889, Ishikawa
  - Site Reference ID/Investigator# 42768, Ishikawa
  - Site Reference ID/Investigator# 58563, Ishikawa
  - Site Reference ID/Investigator# 58600, Ishikawa
  - Site Reference ID/Investigator# 58857, Ishikawa
  - Site Reference ID/Investigator# 39799, Iwafune
  - Site Reference ID/Investigator# 42894, Iwafune
  - Site Reference ID/Investigator# 36059, Kagawa
  - Site Reference ID/Investigator# 36060, Kagawa
  - Site Reference ID/Investigator# 36248, Kagawa
  - Site Reference ID/Investigator# 36491, Kagawa
  - Site Reference ID/Investigator# 36570, Kagawa
  - Site Reference ID/Investigator# 36683, Kagawa
  - Site Reference ID/Investigator# 36687, Kagawa
  - Site Reference ID/Investigator# 36834, Kagawa
  - Site Reference ID/Investigator# 36835, Kagawa
  - Site Reference ID/Investigator# 39657, Kagawa
  - Site Reference ID/Investigator# 39658, Kagawa
  - Site Reference ID/Investigator# 39659, Kagawa
  - Site Reference ID/Investigator# 39660, Kagawa
  - Site Reference ID/Investigator# 39662, Kagawa
  - Site Reference ID/Investigator# 39663, Kagawa
  - Site Reference ID/Investigator# 39664, Kagawa
  - Site Reference ID/Investigator# 39665, Kagawa
  - Site Reference ID/Investigator# 42777, Kagawa
  - Site Reference ID/Investigator# 42814, Kagawa
  - Site Reference ID/Investigator# 58810, Kagawa
  - Site Reference ID/Investigator# 36233, Kagoshima
  - Site Reference ID/Investigator# 36746, Kagoshima
  - Site Reference ID/Investigator# 39661, Kagoshima
  - Site Reference ID/Investigator# 39674, Kagoshima
  - Site Reference ID/Investigator# 39675, Kagoshima
  - Site Reference ID/Investigator# 39676, Kagoshima
  - Site Reference ID/Investigator# 39677, Kagoshima
  - Site Reference ID/Investigator# 39678, Kagoshima
  - Site Reference ID/Investigator# 39679, Kagoshima
  - Site Reference ID/Investigator# 39680, Kagoshima
  - Site Reference ID/Investigator# 39681, Kagoshima
  - Site Reference ID/Investigator# 39682, Kagoshima
  - Site Reference ID/Investigator# 39683, Kagoshima
  - Site Reference ID/Investigator# 39685, Kagoshima
  - Site Reference ID/Investigator# 39688, Kagoshima
  - Site Reference ID/Investigator# 42811, Kagoshima
  - Site Reference ID/Investigator# 42812, Kagoshima
  - Site Reference ID/Investigator# 42813, Kagoshima
  - Site Reference ID/Investigator# 58555, Kagoshima
  - Site Reference ID/Investigator# 58557, Kagoshima
  - Site Reference ID/Investigator# 58560, Kagoshima
  - Site Reference ID/Investigator# 36234, Kanagawa
  - Site Reference ID/Investigator# 36235, Kanagawa
  - Site Reference ID/Investigator# 36236, Kanagawa
  - Site Reference ID/Investigator# 36237, Kanagawa
  - Site Reference ID/Investigator# 36238, Kanagawa
  - Site Reference ID/Investigator# 36240, Kanagawa
  - Site Reference ID/Investigator# 36241, Kanagawa
  - Site Reference ID/Investigator# 36242, Kanagawa
  - Site Reference ID/Investigator# 36243, Kanagawa
  - Site Reference ID/Investigator# 36244, Kanagawa
  - Site Reference ID/Investigator# 36245, Kanagawa
  - Site Reference ID/Investigator# 36246, Kanagawa
  - Site Reference ID/Investigator# 36247, Kanagawa
  - Site Reference ID/Investigator# 36450, Kanagawa
  - Site Reference ID/Investigator# 36545, Kanagawa
  - Site Reference ID/Investigator# 36569, Kanagawa
  - Site Reference ID/Investigator# 36602, Kanagawa
  - Site Reference ID/Investigator# 36654, Kanagawa
  - Site Reference ID/Investigator# 36656, Kanagawa
  - Site Reference ID/Investigator# 36701, Kanagawa
  - Site Reference ID/Investigator# 36790, Kanagawa
  - Site Reference ID/Investigator# 36820, Kanagawa
  - Site Reference ID/Investigator# 36829, Kanagawa
  - Site Reference ID/Investigator# 36837, Kanagawa
  - Site Reference ID/Investigator# 36869, Kanagawa
  - Site Reference ID/Investigator# 36873, Kanagawa
  - Site Reference ID/Investigator# 39684, Kanagawa
  - Site Reference ID/Investigator# 39686, Kanagawa
  - Site Reference ID/Investigator# 39687, Kanagawa
  - Site Reference ID/Investigator# 39689, Kanagawa
  - Site Reference ID/Investigator# 39690, Kanagawa
  - Site Reference ID/Investigator# 39691, Kanagawa
  - Site Reference ID/Investigator# 39694, Kanagawa
  - Site Reference ID/Investigator# 39695, Kanagawa
  - Site Reference ID/Investigator# 39696, Kanagawa
  - Site Reference ID/Investigator# 39698, Kanagawa
  - Site Reference ID/Investigator# 39699, Kanagawa
  - Site Reference ID/Investigator# 39700, Kanagawa
  - Site Reference ID/Investigator# 39705, Kanagawa
  - Site Reference ID/Investigator# 39707, Kanagawa
  - Site Reference ID/Investigator# 39708, Kanagawa
  - Site Reference ID/Investigator# 39709, Kanagawa
  - Site Reference ID/Investigator# 39710, Kanagawa
  - Site Reference ID/Investigator# 39711, Kanagawa
  - Site Reference ID/Investigator# 39712, Kanagawa
  - Site Reference ID/Investigator# 39713, Kanagawa
  - Site Reference ID/Investigator# 39714, Kanagawa
  - Site Reference ID/Investigator# 39716, Kanagawa
  - Site Reference ID/Investigator# 39717, Kanagawa
  - Site Reference ID/Investigator# 39718, Kanagawa
  - Site Reference ID/Investigator# 39720, Kanagawa
  - Site Reference ID/Investigator# 39722, Kanagawa
  - Site Reference ID/Investigator# 39723, Kanagawa
  - Site Reference ID/Investigator# 39724, Kanagawa
  - Site Reference ID/Investigator# 39725, Kanagawa
  - Site Reference ID/Investigator# 42736, Kanagawa
  - Site Reference ID/Investigator# 42822, Kanagawa
  - Site Reference ID/Investigator# 42823, Kanagawa
  - Site Reference ID/Investigator# 42824, Kanagawa
  - Site Reference ID/Investigator# 42826, Kanagawa
  - Site Reference ID/Investigator# 42827, Kanagawa
  - Site Reference ID/Investigator# 58546, Kanagawa
  - Site Reference ID/Investigator# 58549, Kanagawa
  - Site Reference ID/Investigator# 58564, Kanagawa
  - Site Reference ID/Investigator# 58573, Kanagawa
  - Site Reference ID/Investigator# 58574, Kanagawa
  - Site Reference ID/Investigator# 58677, Kanagawa
  - Site Reference ID/Investigator# 58678, Kanagawa
  - Site Reference ID/Investigator# 58679, Kanagawa
  - Site Reference ID/Investigator# 58788, Kanagawa
  - Site Reference ID/Investigator# 58791, Kanagawa
  - Site Reference ID/Investigator# 58796, Kanagawa
  - Site Reference ID/Investigator# 58806, Kanagawa
  - Site Reference ID/Investigator# 58835, Kanagawa
  - Site Reference ID/Investigator# 58836, Kanagawa
  - Site Reference ID/Investigator# 58837, Kanagawa
  - Site Reference ID/Investigator# 58870, Kanagawa
  - Site Reference ID/Investigator# 36846, Kanazawa
  - Site Reference ID/Investigator# 39645, Kanazawa
  - Site Reference ID/Investigator# 39646, Kanazawa
  - Site Reference ID/Investigator# 39647, Kanazawa
  - Site Reference ID/Investigator# 39886, Kanazawa
  - Site Reference ID/Investigator# 36836, Kashihara
  - Site Reference ID/Investigator# 36844, Kashihara
  - Site Reference ID/Investigator# 36941, Kashihara
  - Site Reference ID/Investigator# 36743, Kasugai
  - Site Reference ID/Investigator# 39453, Kawagow
  - Site Reference ID/Investigator# 39706, Kawasaki
  - Site Reference ID/Investigator# 39817, Kawasaki
  - Site Reference ID/Investigator# 58550, Kawasaki
  - Site Reference ID/Investigator# 36946, Kitakami
  - Site Reference ID/Investigator# 36668, Kitakyushu
  - Site Reference ID/Investigator# 36913, Kitakyushu
  - Site Reference ID/Investigator# 39536, Kobe
  - Site Reference ID/Investigator# 39544, Kobe
  - Site Reference ID/Investigator# 36249, Kochi
  - Site Reference ID/Investigator# 36467, Kochi
  - Site Reference ID/Investigator# 36589, Kochi
  - Site Reference ID/Investigator# 36731, Kochi
  - Site Reference ID/Investigator# 36732, Kochi
  - Site Reference ID/Investigator# 36745, Kochi
  - Site Reference ID/Investigator# 36789, Kochi
  - Site Reference ID/Investigator# 39719, Kochi
  - Site Reference ID/Investigator# 39721, Kochi
  - Site Reference ID/Investigator# 39742, Kochi
  - Site Reference ID/Investigator# 39743, Kochi
  - Site Reference ID/Investigator# 39747, Kochi
  - Site Reference ID/Investigator# 39748, Kochi
  - Site Reference ID/Investigator# 42819, Kochi
  - Site Reference ID/Investigator# 42820, Kochi
  - Site Reference ID/Investigator# 42821, Kochi
  - Site Reference ID/Investigator# 58551, Kochi
  - Site Reference ID/Investigator# 58866, Kochi
  - Site Reference ID/Investigator# 36250, Kumamoto
  - Site Reference ID/Investigator# 36251, Kumamoto
  - Site Reference ID/Investigator# 36547, Kumamoto
  - Site Reference ID/Investigator# 36586, Kumamoto
  - Site Reference ID/Investigator# 36669, Kumamoto
  - Site Reference ID/Investigator# 36700, Kumamoto
  - Site Reference ID/Investigator# 39744, Kumamoto
  - Site Reference ID/Investigator# 39745, Kumamoto
  - Site Reference ID/Investigator# 39746, Kumamoto
  - Site Reference ID/Investigator# 39749, Kumamoto
  - Site Reference ID/Investigator# 39750, Kumamoto
  - Site Reference ID/Investigator# 39753, Kumamoto
  - Site Reference ID/Investigator# 39756, Kumamoto
  - Site Reference ID/Investigator# 42746, Kumamoto
  - Site Reference ID/Investigator# 42810, Kumamoto
  - Site Reference ID/Investigator# 42892, Kumamoto
  - Site Reference ID/Investigator# 58556, Kumamoto
  - Site Reference ID/Investigator# 58559, Kumamoto
  - Site Reference ID/Investigator# 36119, Kurume
  - Site Reference ID/Investigator# 36252, Kyoto
  - Site Reference ID/Investigator# 36253, Kyoto
  - Site Reference ID/Investigator# 36254, Kyoto
  - Site Reference ID/Investigator# 36255, Kyoto
  - Site Reference ID/Investigator# 36256, Kyoto
  - Site Reference ID/Investigator# 36257, Kyoto
  - Site Reference ID/Investigator# 36258, Kyoto
  - Site Reference ID/Investigator# 36259, Kyoto
  - Site Reference ID/Investigator# 36679, Kyoto
  - Site Reference ID/Investigator# 36697, Kyoto
  - Site Reference ID/Investigator# 36740, Kyoto
  - Site Reference ID/Investigator# 36921, Kyoto
  - Site Reference ID/Investigator# 36953, Kyoto
  - Site Reference ID/Investigator# 39127, Kyoto
  - Site Reference ID/Investigator# 39751, Kyoto
  - Site Reference ID/Investigator# 39752, Kyoto
  - Site Reference ID/Investigator# 39754, Kyoto
  - Site Reference ID/Investigator# 39755, Kyoto
  - Site Reference ID/Investigator# 39757, Kyoto
  - Site Reference ID/Investigator# 39758, Kyoto
  - Site Reference ID/Investigator# 39759, Kyoto
  - Site Reference ID/Investigator# 39760, Kyoto
  - Site Reference ID/Investigator# 39761, Kyoto
  - Site Reference ID/Investigator# 39763, Kyoto
  - Site Reference ID/Investigator# 39764, Kyoto
  - Site Reference ID/Investigator# 39767, Kyoto
  - Site Reference ID/Investigator# 39768, Kyoto
  - Site Reference ID/Investigator# 42726, Kyoto
  - Site Reference ID/Investigator# 42748, Kyoto
  - Site Reference ID/Investigator# 42750, Kyoto
  - Site Reference ID/Investigator# 42752, Kyoto
  - Site Reference ID/Investigator# 42774, Kyoto
  - Site Reference ID/Investigator# 42776, Kyoto
  - Site Reference ID/Investigator# 42779, Kyoto
  - Site Reference ID/Investigator# 42802, Kyoto
  - Site Reference ID/Investigator# 42890, Kyoto
  - Site Reference ID/Investigator# 42913, Kyoto
  - Site Reference ID/Investigator# 42922, Kyoto
  - Site Reference ID/Investigator# 42923, Kyoto
  - Site Reference ID/Investigator# 42925, Kyoto
  - Site Reference ID/Investigator# 58554, Kyoto
  - Site Reference ID/Investigator# 58577, Kyoto
  - Site Reference ID/Investigator# 58613, Kyoto
  - Site Reference ID/Investigator# 58707, Kyoto
  - Site Reference ID/Investigator# 58708, Kyoto
  - Site Reference ID/Investigator# 58709, Kyoto
  - Site Reference ID/Investigator# 58710, Kyoto
  - Site Reference ID/Investigator# 58711, Kyoto
  - Site Reference ID/Investigator# 58712, Kyoto
  - Site Reference ID/Investigator# 58797, Kyoto
  - Site Reference ID/Investigator# 58858, Kyoto
  - Site Reference ID/Investigator# 58859, Kyoto
  - Site Reference ID/Investigator# 39492, Maebashi
  - Site Reference ID/Investigator# 58715, Matsuyama
  - Site Reference ID/Investigator# 36260, Mie
  - Site Reference ID/Investigator# 36468, Mie
  - Site Reference ID/Investigator# 36599, Mie
  - Site Reference ID/Investigator# 36729, Mie
  - Site Reference ID/Investigator# 36798, Mie
  - Site Reference ID/Investigator# 36949, Mie
  - Site Reference ID/Investigator# 36950, Mie
  - Site Reference ID/Investigator# 39259, Mie
  - Site Reference ID/Investigator# 39302, Mie
  - Site Reference ID/Investigator# 39303, Mie
  - Site Reference ID/Investigator# 39304, Mie
  - Site Reference ID/Investigator# 39306, Mie
  - Site Reference ID/Investigator# 39309, Mie
  - Site Reference ID/Investigator# 39762, Mie
  - Site Reference ID/Investigator# 39765, Mie
  - Site Reference ID/Investigator# 42859, Mie
  - Site Reference ID/Investigator# 58584, Mie
  - Site Reference ID/Investigator# 58591, Mie
  - Site Reference ID/Investigator# 58594, Mie
  - Site Reference ID/Investigator# 58692, Mie
  - Site Reference ID/Investigator# 58793, Mie
  - Site Reference ID/Investigator# 36261, Miyagi
  - Site Reference ID/Investigator# 36262, Miyagi
  - Site Reference ID/Investigator# 36263, Miyagi
  - Site Reference ID/Investigator# 36264, Miyagi
  - Site Reference ID/Investigator# 36265, Miyagi
  - Site Reference ID/Investigator# 36665, Miyagi
  - Site Reference ID/Investigator# 36793, Miyagi
  - Site Reference ID/Investigator# 36802, Miyagi
  - Site Reference ID/Investigator# 36824, Miyagi
  - Site Reference ID/Investigator# 39305, Miyagi
  - Site Reference ID/Investigator# 39307, Miyagi
  - Site Reference ID/Investigator# 39311, Miyagi
  - Site Reference ID/Investigator# 39312, Miyagi
  - Site Reference ID/Investigator# 39314, Miyagi
  - Site Reference ID/Investigator# 39316, Miyagi
  - Site Reference ID/Investigator# 39318, Miyagi
  - Site Reference ID/Investigator# 39917, Miyagi
  - Site Reference ID/Investigator# 42775, Miyagi
  - Site Reference ID/Investigator# 42780, Miyagi
  - Site Reference ID/Investigator# 42943, Miyagi
  - Site Reference ID/Investigator# 58552, Miyagi
  - Site Reference ID/Investigator# 36266, Miyazaki
  - Site Reference ID/Investigator# 36267, Miyazaki
  - Site Reference ID/Investigator# 36268, Miyazaki
  - Site Reference ID/Investigator# 36270, Miyazaki
  - Site Reference ID/Investigator# 36271, Miyazaki
  - Site Reference ID/Investigator# 36272, Miyazaki
  - Site Reference ID/Investigator# 36273, Miyazaki
  - Site Reference ID/Investigator# 36274, Miyazaki
  - Site Reference ID/Investigator# 36559, Miyazaki
  - Site Reference ID/Investigator# 38523, Miyazaki
  - Site Reference ID/Investigator# 39313, Miyazaki
  - Site Reference ID/Investigator# 39319, Miyazaki
  - Site Reference ID/Investigator# 39323, Miyazaki
  - Site Reference ID/Investigator# 39326, Miyazaki
  - Site Reference ID/Investigator# 42809, Miyazaki
  - Site Reference ID/Investigator# 42886, Miyazaki
  - Site Reference ID/Investigator# 58780, Miyazaki
  - Site Reference ID/Investigator# 58781, Miyazaki
  - Site Reference ID/Investigator# 58794, Miyazaki
  - Site Reference ID/Investigator# 58815, Miyazaki
  - Site Reference ID/Investigator# 36275, Nagano
  - Site Reference ID/Investigator# 36276, Nagano
  - Site Reference ID/Investigator# 36277, Nagano
  - Site Reference ID/Investigator# 36278, Nagano
  - Site Reference ID/Investigator# 36279, Nagano
  - Site Reference ID/Investigator# 36280, Nagano
  - Site Reference ID/Investigator# 36281, Nagano
  - Site Reference ID/Investigator# 36282, Nagano
  - Site Reference ID/Investigator# 36283, Nagano
  - Site Reference ID/Investigator# 36284, Nagano
  - Site Reference ID/Investigator# 36515, Nagano
  - Site Reference ID/Investigator# 36551, Nagano
  - Site Reference ID/Investigator# 36556, Nagano
  - Site Reference ID/Investigator# 36603, Nagano
  - Site Reference ID/Investigator# 39320, Nagano
  - Site Reference ID/Investigator# 39321, Nagano
  - Site Reference ID/Investigator# 39322, Nagano
  - Site Reference ID/Investigator# 39324, Nagano
  - Site Reference ID/Investigator# 39327, Nagano
  - Site Reference ID/Investigator# 39328, Nagano
  - Site Reference ID/Investigator# 42897, Nagano
  - Site Reference ID/Investigator# 42911, Nagano
  - Site Reference ID/Investigator# 58565, Nagano
  - Site Reference ID/Investigator# 58571, Nagano
  - Site Reference ID/Investigator# 58658, Nagano
  - Site Reference ID/Investigator# 58803, Nagano
  - Site Reference ID/Investigator# 36285, Nagasaki
  - Site Reference ID/Investigator# 36286, Nagasaki
  - Site Reference ID/Investigator# 36287, Nagasaki
  - Site Reference ID/Investigator# 36288, Nagasaki
  - Site Reference ID/Investigator# 36289, Nagasaki
  - Site Reference ID/Investigator# 36554, Nagasaki
  - Site Reference ID/Investigator# 36728, Nagasaki
  - Site Reference ID/Investigator# 39329, Nagasaki
  - Site Reference ID/Investigator# 39330, Nagasaki
  - Site Reference ID/Investigator# 39331, Nagasaki
  - Site Reference ID/Investigator# 39332, Nagasaki
  - Site Reference ID/Investigator# 39333, Nagasaki
  - Site Reference ID/Investigator# 39334, Nagasaki
  - Site Reference ID/Investigator# 39335, Nagasaki
  - Site Reference ID/Investigator# 39336, Nagasaki
  - Site Reference ID/Investigator# 39337, Nagasaki
  - Site Reference ID/Investigator# 39918, Nagasaki
  - Site Reference ID/Investigator# 58558, Nagasaki
  - Site Reference ID/Investigator# 35910, Nagoya
  - Site Reference ID/Investigator# 35911, Nagoya
  - Site Reference ID/Investigator# 39139, Nagoya
  - Site Reference ID/Investigator# 36290, Nara
  - Site Reference ID/Investigator# 36291, Nara
  - Site Reference ID/Investigator# 36572, Nara
  - Site Reference ID/Investigator# 36574, Nara
  - Site Reference ID/Investigator# 36591, Nara
  - Site Reference ID/Investigator# 36648, Nara
  - Site Reference ID/Investigator# 39338, Nara
  - Site Reference ID/Investigator# 39342, Nara
  - Site Reference ID/Investigator# 39343, Nara
  - Site Reference ID/Investigator# 39344, Nara
  - Site Reference ID/Investigator# 39345, Nara
  - Site Reference ID/Investigator# 39346, Nara
  - Site Reference ID/Investigator# 42781, Nara
  - Site Reference ID/Investigator# 42782, Nara
  - Site Reference ID/Investigator# 42909, Nara
  - Site Reference ID/Investigator# 58702, Nara
  - Site Reference ID/Investigator# 58703, Nara
  - Site Reference ID/Investigator# 58784, Nara
  - Site Reference ID/Investigator# 58853, Nara
  - Site Reference ID/Investigator# 36680, Neyagawa
  - Site Reference ID/Investigator# 42895, Nigata-honmachi
  - Site Reference ID/Investigator# 42901, Nigata-honmachi
  - Site Reference ID/Investigator# 42902, Nigata-honmachi
  - Site Reference ID/Investigator# 36190, Niigata
  - Site Reference ID/Investigator# 36292, Niigata
  - Site Reference ID/Investigator# 36293, Niigata
  - Site Reference ID/Investigator# 36457, Niigata
  - Site Reference ID/Investigator# 36871, Niigata
  - Site Reference ID/Investigator# 36872, Niigata
  - Site Reference ID/Investigator# 36962, Niigata
  - Site Reference ID/Investigator# 39339, Niigata
  - Site Reference ID/Investigator# 39340, Niigata
  - Site Reference ID/Investigator# 39341, Niigata
  - Site Reference ID/Investigator# 39347, Niigata
  - Site Reference ID/Investigator# 39352, Niigata
  - Site Reference ID/Investigator# 39355, Niigata
  - Site Reference ID/Investigator# 42778, Niigata
  - Site Reference ID/Investigator# 58596, Niigata
  - Site Reference ID/Investigator# 39864, Nishinomiya
  - Site Reference ID/Investigator# 36062, Numakunai
  - Site Reference ID/Investigator# 36520, Numakunai
  - Site Reference ID/Investigator# 36736, Numakunai
  - Site Reference ID/Investigator# 36737, Numakunai
  - Site Reference ID/Investigator# 36749, Numakunai
  - Site Reference ID/Investigator# 36932, Numakunai
  - Site Reference ID/Investigator# 39649, Numakunai
  - Site Reference ID/Investigator# 39650, Numakunai
  - Site Reference ID/Investigator# 39652, Numakunai
  - Site Reference ID/Investigator# 39654, Numakunai
  - Site Reference ID/Investigator# 39656, Numakunai
  - Site Reference ID/Investigator# 42869, Numakunai
  - Site Reference ID/Investigator# 42870, Numakunai
  - Site Reference ID/Investigator# 39526, Obihiro
  - Site Reference ID/Investigator# 36183, Okayama
  - Site Reference ID/Investigator# 36185, Okayama
  - Site Reference ID/Investigator# 36186, Okayama
  - Site Reference ID/Investigator# 36188, Okayama
  - Site Reference ID/Investigator# 36558, Okayama
  - Site Reference ID/Investigator# 36671, Okayama
  - Site Reference ID/Investigator# 36795, Okayama
  - Site Reference ID/Investigator# 36875, Okayama
  - Site Reference ID/Investigator# 36931, Okayama
  - Site Reference ID/Investigator# 39356, Okayama
  - Site Reference ID/Investigator# 39359, Okayama
  - Site Reference ID/Investigator# 39360, Okayama
  - Site Reference ID/Investigator# 39361, Okayama
  - Site Reference ID/Investigator# 39362, Okayama
  - Site Reference ID/Investigator# 39363, Okayama
  - Site Reference ID/Investigator# 39364, Okayama
  - Site Reference ID/Investigator# 42788, Okayama
  - Site Reference ID/Investigator# 42838, Okayama
  - Site Reference ID/Investigator# 42840, Okayama
  - Site Reference ID/Investigator# 58566, Okayama
  - Site Reference ID/Investigator# 58860, Okayama
  - Site Reference ID/Investigator# 58874, Okayama
  - Site Reference ID/Investigator# 36613, Okinawa
  - Site Reference ID/Investigator# 36741, Okinawa
  - Site Reference ID/Investigator# 36926, Okinawa
  - Site Reference ID/Investigator# 39365, Okinawa
  - Site Reference ID/Investigator# 39368, Okinawa
  - Site Reference ID/Investigator# 39372, Okinawa
  - Site Reference ID/Investigator# 39373, Okinawa
  - Site Reference ID/Investigator# 39915, Okinawa
  - Site Reference ID/Investigator# 58547, Okinawa
  - Site Reference ID/Investigator# 58608, Okinawa
  - Site Ref # / Investigator 36232, Osaka
  - Site Reference ID/Investigator# 36191, Osaka
  - Site Reference ID/Investigator# 36192, Osaka
  - Site Reference ID/Investigator# 36193, Osaka
  - Site Reference ID/Investigator# 36194, Osaka
  - Site Reference ID/Investigator# 36195, Osaka
  - Site Reference ID/Investigator# 36196, Osaka
  - Site Reference ID/Investigator# 36197, Osaka
  - Site Reference ID/Investigator# 36198, Osaka
  - Site Reference ID/Investigator# 36199, Osaka
  - Site Reference ID/Investigator# 36200, Osaka
  - Site Reference ID/Investigator# 36201, Osaka
  - Site Reference ID/Investigator# 36204, Osaka
  - Site Reference ID/Investigator# 36205, Osaka
  - Site Reference ID/Investigator# 36206, Osaka
  - Site Reference ID/Investigator# 36207, Osaka
  - Site Reference ID/Investigator# 36208, Osaka
  - Site Reference ID/Investigator# 36444, Osaka
  - Site Reference ID/Investigator# 36514, Osaka
  - Site Reference ID/Investigator# 36552, Osaka
  - Site Reference ID/Investigator# 36555, Osaka
  - Site Reference ID/Investigator# 36557, Osaka
  - Site Reference ID/Investigator# 36573, Osaka
  - Site Reference ID/Investigator# 36576, Osaka
  - Site Reference ID/Investigator# 36580, Osaka
  - Site Reference ID/Investigator# 36582, Osaka
  - Site Reference ID/Investigator# 36584, Osaka
  - Site Reference ID/Investigator# 36585, Osaka
  - Site Reference ID/Investigator# 36587, Osaka
  - Site Reference ID/Investigator# 36588, Osaka
  - Site Reference ID/Investigator# 36598, Osaka
  - Site Reference ID/Investigator# 36616, Osaka
  - Site Reference ID/Investigator# 36657, Osaka
  - Site Reference ID/Investigator# 36658, Osaka
  - Site Reference ID/Investigator# 36674, Osaka
  - Site Reference ID/Investigator# 36688, Osaka
  - Site Reference ID/Investigator# 36738, Osaka
  - Site Reference ID/Investigator# 36739, Osaka
  - Site Reference ID/Investigator# 36800, Osaka
  - Site Reference ID/Investigator# 36811, Osaka
  - Site Reference ID/Investigator# 36838, Osaka
  - Site Reference ID/Investigator# 36878, Osaka
  - Site Reference ID/Investigator# 36879, Osaka
  - Site Reference ID/Investigator# 36920, Osaka
  - Site Reference ID/Investigator# 36924, Osaka
  - Site Reference ID/Investigator# 36947, Osaka
  - Site Reference ID/Investigator# 36954, Osaka
  - Site Reference ID/Investigator# 36957, Osaka
  - Site Reference ID/Investigator# 39366, Osaka
  - Site Reference ID/Investigator# 39367, Osaka
  - Site Reference ID/Investigator# 39369, Osaka
  - Site Reference ID/Investigator# 39370, Osaka
  - Site Reference ID/Investigator# 39371, Osaka
  - Site Reference ID/Investigator# 39374, Osaka
  - Site Reference ID/Investigator# 39375, Osaka
  - Site Reference ID/Investigator# 39376, Osaka
  - Site Reference ID/Investigator# 39377, Osaka
  - Site Reference ID/Investigator# 39378, Osaka
  - Site Reference ID/Investigator# 39379, Osaka
  - Site Reference ID/Investigator# 39380, Osaka
  - Site Reference ID/Investigator# 39381, Osaka
  - Site Reference ID/Investigator# 39382, Osaka
  - Site Reference ID/Investigator# 39383, Osaka
  - Site Reference ID/Investigator# 39384, Osaka
  - Site Reference ID/Investigator# 39385, Osaka
  - Site Reference ID/Investigator# 39386, Osaka
  - Site Reference ID/Investigator# 39387, Osaka
  - Site Reference ID/Investigator# 39388, Osaka
  - Site Reference ID/Investigator# 39389, Osaka
  - Site Reference ID/Investigator# 39390, Osaka
  - Site Reference ID/Investigator# 39391, Osaka
  - Site Reference ID/Investigator# 39392, Osaka
  - Site Reference ID/Investigator# 39393, Osaka
  - Site Reference ID/Investigator# 39394, Osaka
  - Site Reference ID/Investigator# 39395, Osaka
  - Site Reference ID/Investigator# 39396, Osaka
  - Site Reference ID/Investigator# 39397, Osaka
  - Site Reference ID/Investigator# 39398, Osaka
  - Site Reference ID/Investigator# 39399, Osaka
  - Site Reference ID/Investigator# 39400, Osaka
  - Site Reference ID/Investigator# 39401, Osaka
  - Site Reference ID/Investigator# 39402, Osaka
  - Site Reference ID/Investigator# 39404, Osaka
  - Site Reference ID/Investigator# 39407, Osaka
  - Site Reference ID/Investigator# 39408, Osaka
  - Site Reference ID/Investigator# 39409, Osaka
  - Site Reference ID/Investigator# 39410, Osaka
  - Site Reference ID/Investigator# 39411, Osaka
  - Site Reference ID/Investigator# 39412, Osaka
  - Site Reference ID/Investigator# 39413, Osaka
  - Site Reference ID/Investigator# 39414, Osaka
  - Site Reference ID/Investigator# 39415, Osaka
  - Site Reference ID/Investigator# 39416, Osaka
  - Site Reference ID/Investigator# 39417, Osaka
  - Site Reference ID/Investigator# 39418, Osaka
  - Site Reference ID/Investigator# 39419, Osaka
  - Site Reference ID/Investigator# 39421, Osaka
  - Site Reference ID/Investigator# 39422, Osaka
  - Site Reference ID/Investigator# 39423, Osaka
  - Site Reference ID/Investigator# 39425, Osaka
  - Site Reference ID/Investigator# 39426, Osaka
  - Site Reference ID/Investigator# 39912, Osaka
  - Site Reference ID/Investigator# 39913, Osaka
  - Site Reference ID/Investigator# 39914, Osaka
  - Site Reference ID/Investigator# 42716, Osaka
  - Site Reference ID/Investigator# 42730, Osaka
  - Site Reference ID/Investigator# 42745, Osaka
  - Site Reference ID/Investigator# 42751, Osaka
  - Site Reference ID/Investigator# 42755, Osaka
  - Site Reference ID/Investigator# 42789, Osaka
  - Site Reference ID/Investigator# 42790, Osaka
  - Site Reference ID/Investigator# 42791, Osaka
  - Site Reference ID/Investigator# 42887, Osaka
  - Site Reference ID/Investigator# 42904, Osaka
  - Site Reference ID/Investigator# 42905, Osaka
  - Site Reference ID/Investigator# 42907, Osaka
  - Site Reference ID/Investigator# 42908, Osaka
  - Site Reference ID/Investigator# 42910, Osaka
  - Site Reference ID/Investigator# 42912, Osaka
  - Site Reference ID/Investigator# 42914, Osaka
  - Site Reference ID/Investigator# 42915, Osaka
  - Site Reference ID/Investigator# 42916, Osaka
  - Site Reference ID/Investigator# 42917, Osaka
  - Site Reference ID/Investigator# 42918, Osaka
  - Site Reference ID/Investigator# 42919, Osaka
  - Site Reference ID/Investigator# 42920, Osaka
  - Site Reference ID/Investigator# 42921, Osaka
  - Site Reference ID/Investigator# 42926, Osaka
  - Site Reference ID/Investigator# 42928, Osaka
  - Site Reference ID/Investigator# 42929, Osaka
  - Site Reference ID/Investigator# 58553, Osaka
  - Site Reference ID/Investigator# 58575, Osaka
  - Site Reference ID/Investigator# 58576, Osaka
  - Site Reference ID/Investigator# 58582, Osaka
  - Site Reference ID/Investigator# 58585, Osaka
  - Site Reference ID/Investigator# 58588, Osaka
  - Site Reference ID/Investigator# 58602, Osaka
  - Site Reference ID/Investigator# 58603, Osaka
  - Site Reference ID/Investigator# 58604, Osaka
  - Site Reference ID/Investigator# 58694, Osaka
  - Site Reference ID/Investigator# 58695, Osaka
  - Site Reference ID/Investigator# 58696, Osaka
  - Site Reference ID/Investigator# 58697, Osaka
  - Site Reference ID/Investigator# 58698, Osaka
  - Site Reference ID/Investigator# 58699, Osaka
  - Site Reference ID/Investigator# 58700, Osaka
  - Site Reference ID/Investigator# 58701, Osaka
  - Site Reference ID/Investigator# 58795, Osaka
  - Site Reference ID/Investigator# 58805, Osaka
  - Site Reference ID/Investigator# 58816, Osaka
  - Site Reference ID/Investigator# 58851, Osaka
  - Site Reference ID/Investigator# 58852, Osaka
  - Site Reference ID/Investigator# 58871, Osaka
  - Site Reference ID/Investigator# 36182, Ōita
  - Site Reference ID/Investigator# 36184, Ōita
  - Site Reference ID/Investigator# 36187, Ōita
  - Site Reference ID/Investigator# 36189, Ōita
  - Site Reference ID/Investigator# 36567, Ōita
  - Site Reference ID/Investigator# 36809, Ōita
  - Site Reference ID/Investigator# 36815, Ōita
  - Site Reference ID/Investigator# 36825, Ōita
  - Site Reference ID/Investigator# 36826, Ōita
  - Site Reference ID/Investigator# 36905, Ōita
  - Site Reference ID/Investigator# 39348, Ōita
  - Site Reference ID/Investigator# 39349, Ōita
  - Site Reference ID/Investigator# 39350, Ōita
  - Site Reference ID/Investigator# 39351, Ōita
  - Site Reference ID/Investigator# 39353, Ōita
  - Site Reference ID/Investigator# 39354, Ōita
  - Site Reference ID/Investigator# 42724, Ōita
  - Site Reference ID/Investigator# 42785, Ōita
  - Site Reference ID/Investigator# 42808, Ōita
  - Site Reference ID/Investigator# 58586, Ōita
  - Site Reference ID/Investigator# 39315, Ōsaki
  - Site Reference ID/Investigator# 42942, Ōsaki
  - Site Reference ID/Investigator# 36203, Saga
  - Site Reference ID/Investigator# 39420, Saga
  - Site Reference ID/Investigator# 39424, Saga
  - Site Reference ID/Investigator# 39427, Saga
  - Site Reference ID/Investigator# 42806, Saga
  - Site Reference ID/Investigator# 42807, Saga
  - Site Reference ID/Investigator# 58869, Saga
  - Site Reference ID/Investigator# 36202, Saitama
  - Site Reference ID/Investigator# 36209, Saitama
  - Site Reference ID/Investigator# 36210, Saitama
  - Site Reference ID/Investigator# 36211, Saitama
  - Site Reference ID/Investigator# 36212, Saitama
  - Site Reference ID/Investigator# 36213, Saitama
  - Site Reference ID/Investigator# 36214, Saitama
  - Site Reference ID/Investigator# 36215, Saitama
  - Site Reference ID/Investigator# 36216, Saitama
  - Site Reference ID/Investigator# 36217, Saitama
  - Site Reference ID/Investigator# 36219, Saitama
  - Site Reference ID/Investigator# 36220, Saitama
  - Site Reference ID/Investigator# 36446, Saitama
  - Site Reference ID/Investigator# 36456, Saitama
  - Site Reference ID/Investigator# 36469, Saitama
  - Site Reference ID/Investigator# 36479, Saitama
  - Site Reference ID/Investigator# 36646, Saitama
  - Site Reference ID/Investigator# 36734, Saitama
  - Site Reference ID/Investigator# 36747, Saitama
  - Site Reference ID/Investigator# 36831, Saitama
  - Site Reference ID/Investigator# 36951, Saitama
  - Site Reference ID/Investigator# 39428, Saitama
  - Site Reference ID/Investigator# 39429, Saitama
  - Site Reference ID/Investigator# 39430, Saitama
  - Site Reference ID/Investigator# 39431, Saitama
  - Site Reference ID/Investigator# 39432, Saitama
  - Site Reference ID/Investigator# 39433, Saitama
  - Site Reference ID/Investigator# 39434, Saitama
  - Site Reference ID/Investigator# 39435, Saitama
  - Site Reference ID/Investigator# 39436, Saitama
  - Site Reference ID/Investigator# 39437, Saitama
  - Site Reference ID/Investigator# 39438, Saitama
  - Site Reference ID/Investigator# 39439, Saitama
  - Site Reference ID/Investigator# 39440, Saitama
  - Site Reference ID/Investigator# 39441, Saitama
  - Site Reference ID/Investigator# 39442, Saitama
  - Site Reference ID/Investigator# 39443, Saitama
  - Site Reference ID/Investigator# 39444, Saitama
  - Site Reference ID/Investigator# 39445, Saitama
  - Site Reference ID/Investigator# 39447, Saitama
  - Site Reference ID/Investigator# 39448, Saitama
  - Site Reference ID/Investigator# 39449, Saitama
  - Site Reference ID/Investigator# 39450, Saitama
  - Site Reference ID/Investigator# 39451, Saitama
  - Site Reference ID/Investigator# 39452, Saitama
  - Site Reference ID/Investigator# 39454, Saitama
  - Site Reference ID/Investigator# 39455, Saitama
  - Site Reference ID/Investigator# 39459, Saitama
  - Site Reference ID/Investigator# 39916, Saitama
  - Site Reference ID/Investigator# 42739, Saitama
  - Site Reference ID/Investigator# 42783, Saitama
  - Site Reference ID/Investigator# 42784, Saitama
  - Site Reference ID/Investigator# 42787, Saitama
  - Site Reference ID/Investigator# 42834, Saitama
  - Site Reference ID/Investigator# 42835, Saitama
  - Site Reference ID/Investigator# 42836, Saitama
  - Site Reference ID/Investigator# 42837, Saitama
  - Site Reference ID/Investigator# 42888, Saitama
  - Site Reference ID/Investigator# 58548, Saitama
  - Site Reference ID/Investigator# 58572, Saitama
  - Site Reference ID/Investigator# 58581, Saitama
  - Site Reference ID/Investigator# 58589, Saitama
  - Site Reference ID/Investigator# 58590, Saitama
  - Site Reference ID/Investigator# 58669, Saitama
  - Site Reference ID/Investigator# 58670, Saitama
  - Site Reference ID/Investigator# 58671, Saitama
  - Site Reference ID/Investigator# 58672, Saitama
  - Site Reference ID/Investigator# 58673, Saitama
  - Site Reference ID/Investigator# 58674, Saitama
  - Site Reference ID/Investigator# 58675, Saitama
  - Site Reference ID/Investigator# 58799, Saitama
  - Site Reference ID/Investigator# 58812, Saitama
  - Site Reference ID/Investigator# 58832, Saitama
  - Site Reference ID/Investigator# 58833, Saitama
  - Site Reference ID/Investigator# 58834, Saitama
  - Site Reference ID/Investigator# 36939, Sayama
  - Site Reference ID/Investigator# 36940, Sayama
  - Site Reference ID/Investigator# 36218, Shiga
  - Site Reference ID/Investigator# 36224, Shiga
  - Site Reference ID/Investigator# 36225, Shiga
  - Site Reference ID/Investigator# 36226, Shiga
  - Site Reference ID/Investigator# 36832, Shiga
  - Site Reference ID/Investigator# 39310, Shiga
  - Site Reference ID/Investigator# 39456, Shiga
  - Site Reference ID/Investigator# 39457, Shiga
  - Site Reference ID/Investigator# 39460, Shiga
  - Site Reference ID/Investigator# 39461, Shiga
  - Site Reference ID/Investigator# 39462, Shiga
  - Site Reference ID/Investigator# 39463, Shiga
  - Site Reference ID/Investigator# 39775, Shiga
  - Site Reference ID/Investigator# 42786, Shiga
  - Site Reference ID/Investigator# 42803, Shiga
  - Site Reference ID/Investigator# 42804, Shiga
  - Site Reference ID/Investigator# 39769, Shimane
  - Site Reference ID/Investigator# 39771, Shimane
  - Site Reference ID/Investigator# 39772, Shimane
  - Site Reference ID/Investigator# 39773, Shimane
  - Site Reference ID/Investigator# 39776, Shimane
  - Site Reference ID/Investigator# 39777, Shimane
  - Site Reference ID/Investigator# 58579, Shimane
  - Site Reference ID/Investigator# 58713, Shimane
  - Site Reference ID/Investigator# 58802, Shimane
  - Site Reference ID/Investigator# 39800, Shimotsuke
  - Site Reference ID/Investigator# 36117, Shizuoka
  - Site Reference ID/Investigator# 36123, Shizuoka
  - Site Reference ID/Investigator# 36126, Shizuoka
  - Site Reference ID/Investigator# 36221, Shizuoka
  - Site Reference ID/Investigator# 36222, Shizuoka
  - Site Reference ID/Investigator# 36223, Shizuoka
  - Site Reference ID/Investigator# 36227, Shizuoka
  - Site Reference ID/Investigator# 36228, Shizuoka
  - Site Reference ID/Investigator# 36229, Shizuoka
  - Site Reference ID/Investigator# 36230, Shizuoka
  - Site Reference ID/Investigator# 36231, Shizuoka
  - Site Reference ID/Investigator# 36480, Shizuoka
  - Site Reference ID/Investigator# 36553, Shizuoka
  - Site Reference ID/Investigator# 36607, Shizuoka
  - Site Reference ID/Investigator# 36609, Shizuoka
  - Site Reference ID/Investigator# 36827, Shizuoka
  - Site Reference ID/Investigator# 36842, Shizuoka
  - Site Reference ID/Investigator# 36877, Shizuoka
  - Site Reference ID/Investigator# 39774, Shizuoka
  - Site Reference ID/Investigator# 39778, Shizuoka
  - Site Reference ID/Investigator# 39779, Shizuoka
  - Site Reference ID/Investigator# 39780, Shizuoka
  - Site Reference ID/Investigator# 39781, Shizuoka
  - Site Reference ID/Investigator# 39782, Shizuoka
  - Site Reference ID/Investigator# 39783, Shizuoka
  - Site Reference ID/Investigator# 39784, Shizuoka
  - Site Reference ID/Investigator# 39785, Shizuoka
  - Site Reference ID/Investigator# 39786, Shizuoka
  - Site Reference ID/Investigator# 39789, Shizuoka
  - Site Reference ID/Investigator# 39790, Shizuoka
  - Site Reference ID/Investigator# 39791, Shizuoka
  - Site Reference ID/Investigator# 39792, Shizuoka
  - Site Reference ID/Investigator# 39793, Shizuoka
  - Site Reference ID/Investigator# 42731, Shizuoka
  - Site Reference ID/Investigator# 42847, Shizuoka
  - Site Reference ID/Investigator# 42848, Shizuoka
  - Site Reference ID/Investigator# 42849, Shizuoka
  - Site Reference ID/Investigator# 42850, Shizuoka
  - Site Reference ID/Investigator# 42889, Shizuoka
  - Site Reference ID/Investigator# 58593, Shizuoka
  - Site Reference ID/Investigator# 58683, Shizuoka
  - Site Reference ID/Investigator# 58684, Shizuoka
  - Site Reference ID/Investigator# 58685, Shizuoka
  - Site Reference ID/Investigator# 58686, Shizuoka
  - Site Reference ID/Investigator# 58693, Shizuoka
  - Site Reference ID/Investigator# 58840, Shizuoka
  - Site Reference ID/Investigator# 58841, Shizuoka
  - Site Reference ID/Investigator# 58842, Shizuoka
  - Site Reference ID/Investigator# 42829, Shība
  - Site Ref # / Investigator 72773, Suwa
  - Site Reference ID/Investigator# 36730, Takamatsu
  - Site Reference ID/Investigator# 39403, Takatsuki
  - Site Reference ID/Investigator# 39405, Takatsuki
  - Site Reference ID/Investigator# 39406, Takatsuki
  - Site Reference ID/Investigator# 36124, Tochigi
  - Site Reference ID/Investigator# 36127, Tochigi
  - Site Reference ID/Investigator# 36128, Tochigi
  - Site Reference ID/Investigator# 36691, Tochigi
  - Site Reference ID/Investigator# 36874, Tochigi
  - Site Reference ID/Investigator# 36876, Tochigi
  - Site Reference ID/Investigator# 36880, Tochigi
  - Site Reference ID/Investigator# 36881, Tochigi
  - Site Reference ID/Investigator# 36882, Tochigi
  - Site Reference ID/Investigator# 36884, Tochigi
  - Site Reference ID/Investigator# 36887, Tochigi
  - Site Reference ID/Investigator# 36888, Tochigi
  - Site Reference ID/Investigator# 36930, Tochigi
  - Site Reference ID/Investigator# 36959, Tochigi
  - Site Reference ID/Investigator# 36960, Tochigi
  - Site Reference ID/Investigator# 36961, Tochigi
  - Site Reference ID/Investigator# 38524, Tochigi
  - Site Reference ID/Investigator# 39787, Tochigi
  - Site Reference ID/Investigator# 39788, Tochigi
  - Site Reference ID/Investigator# 39794, Tochigi
  - Site Reference ID/Investigator# 39795, Tochigi
  - Site Reference ID/Investigator# 39796, Tochigi
  - Site Reference ID/Investigator# 39797, Tochigi
  - Site Reference ID/Investigator# 39798, Tochigi
  - Site Reference ID/Investigator# 39801, Tochigi
  - Site Reference ID/Investigator# 39802, Tochigi
  - Site Reference ID/Investigator# 42727, Tochigi
  - Site Reference ID/Investigator# 42728, Tochigi
  - Site Reference ID/Investigator# 42899, Tochigi
  - Site Reference ID/Investigator# 58544, Tochigi
  - Site Reference ID/Investigator# 58567, Tochigi
  - Site Reference ID/Investigator# 58609, Tochigi
  - Site Reference ID/Investigator# 58655, Tochigi
  - Site Reference ID/Investigator# 58656, Tochigi
  - Site Reference ID/Investigator# 58826, Tochigi
  - Site Reference ID/Investigator# 36125, Tokushima
  - Site Reference ID/Investigator# 36129, Tokushima
  - Site Reference ID/Investigator# 36577, Tokushima
  - Site Reference ID/Investigator# 36685, Tokushima
  - Site Reference ID/Investigator# 36883, Tokushima
  - Site Reference ID/Investigator# 39803, Tokushima
  - Site Reference ID/Investigator# 39806, Tokushima
  - Site Reference ID/Investigator# 39809, Tokushima
  - Site Reference ID/Investigator# 39810, Tokushima
  - Site Reference ID/Investigator# 42747, Tokushima
  - Site Reference ID/Investigator# 42816, Tokushima
  - Site Reference ID/Investigator# 58865, Tokushima
  - Site Reference ID/Investigator# 14581, Tokyo
  - Site Reference ID/Investigator# 36131, Tokyo
  - Site Reference ID/Investigator# 36132, Tokyo
  - Site Reference ID/Investigator# 36133, Tokyo
  - Site Reference ID/Investigator# 36134, Tokyo
  - Site Reference ID/Investigator# 36135, Tokyo
  - Site Reference ID/Investigator# 36136, Tokyo
  - Site Reference ID/Investigator# 36138, Tokyo
  - Site Reference ID/Investigator# 36139, Tokyo
  - Site Reference ID/Investigator# 36140, Tokyo
  - Site Reference ID/Investigator# 36141, Tokyo
  - Site Reference ID/Investigator# 36142, Tokyo
  - Site Reference ID/Investigator# 36143, Tokyo
  - Site Reference ID/Investigator# 36144, Tokyo
  - Site Reference ID/Investigator# 36145, Tokyo
  - Site Reference ID/Investigator# 36146, Tokyo
  - Site Reference ID/Investigator# 36147, Tokyo
  - Site Reference ID/Investigator# 36149, Tokyo
  - Site Reference ID/Investigator# 36150, Tokyo
  - Site Reference ID/Investigator# 36151, Tokyo
  - Site Reference ID/Investigator# 36153, Tokyo
  - Site Reference ID/Investigator# 36154, Tokyo
  - Site Reference ID/Investigator# 36155, Tokyo
  - Site Reference ID/Investigator# 36156, Tokyo
  - Site Reference ID/Investigator# 36157, Tokyo
  - Site Reference ID/Investigator# 36158, Tokyo
  - Site Reference ID/Investigator# 36159, Tokyo
  - Site Reference ID/Investigator# 36160, Tokyo
  - Site Reference ID/Investigator# 36161, Tokyo
  - Site Reference ID/Investigator# 36162, Tokyo
  - Site Reference ID/Investigator# 36163, Tokyo
  - Site Reference ID/Investigator# 36164, Tokyo
  - Site Reference ID/Investigator# 36165, Tokyo
  - Site Reference ID/Investigator# 36166, Tokyo
  - Site Reference ID/Investigator# 36167, Tokyo
  - Site Reference ID/Investigator# 36168, Tokyo
  - Site Reference ID/Investigator# 36169, Tokyo
  - Site Reference ID/Investigator# 36453, Tokyo
  - Site Reference ID/Investigator# 36561, Tokyo
  - Site Reference ID/Investigator# 36562, Tokyo
  - Site Reference ID/Investigator# 36563, Tokyo
  - Site Reference ID/Investigator# 36565, Tokyo
  - Site Reference ID/Investigator# 36575, Tokyo
  - Site Reference ID/Investigator# 36581, Tokyo
  - Site Reference ID/Investigator# 36590, Tokyo
  - Site Reference ID/Investigator# 36593, Tokyo
  - Site Reference ID/Investigator# 36594, Tokyo
  - Site Reference ID/Investigator# 36596, Tokyo
  - Site Reference ID/Investigator# 36615, Tokyo
  - Site Reference ID/Investigator# 36641, Tokyo
  - Site Reference ID/Investigator# 36653, Tokyo
  - Site Reference ID/Investigator# 36664, Tokyo
  - Site Reference ID/Investigator# 36682, Tokyo
  - Site Reference ID/Investigator# 36684, Tokyo
  - Site Reference ID/Investigator# 36690, Tokyo
  - Site Reference ID/Investigator# 36698, Tokyo
  - Site Reference ID/Investigator# 36725, Tokyo
  - Site Reference ID/Investigator# 36726, Tokyo
  - Site Reference ID/Investigator# 36751, Tokyo
  - Site Reference ID/Investigator# 36792, Tokyo
  - Site Reference ID/Investigator# 36794, Tokyo
  - Site Reference ID/Investigator# 36803, Tokyo
  - Site Reference ID/Investigator# 36810, Tokyo
  - Site Reference ID/Investigator# 36812, Tokyo
  - Site Reference ID/Investigator# 36816, Tokyo
  - Site Reference ID/Investigator# 36818, Tokyo
  - Site Reference ID/Investigator# 36845, Tokyo
  - Site Reference ID/Investigator# 36885, Tokyo
  - Site Reference ID/Investigator# 36886, Tokyo
  - Site Reference ID/Investigator# 36915, Tokyo
  - Site Reference ID/Investigator# 36919, Tokyo
  - Site Reference ID/Investigator# 36934, Tokyo
  - Site Reference ID/Investigator# 36956, Tokyo
  - Site Reference ID/Investigator# 36963, Tokyo
  - Site Reference ID/Investigator# 39582, Tokyo
  - Site Reference ID/Investigator# 39583, Tokyo
  - Site Reference ID/Investigator# 39584, Tokyo
  - Site Reference ID/Investigator# 39585, Tokyo
  - Site Reference ID/Investigator# 39622, Tokyo
  - Site Reference ID/Investigator# 39623, Tokyo
  - Site Reference ID/Investigator# 39697, Tokyo
  - Site Reference ID/Investigator# 39804, Tokyo
  - Site Reference ID/Investigator# 39805, Tokyo
  - Site Reference ID/Investigator# 39807, Tokyo
  - Site Reference ID/Investigator# 39808, Tokyo
  - Site Reference ID/Investigator# 39811, Tokyo
  - Site Reference ID/Investigator# 39812, Tokyo
  - Site Reference ID/Investigator# 39813, Tokyo
  - Site Reference ID/Investigator# 39815, Tokyo
  - Site Reference ID/Investigator# 39816, Tokyo
  - Site Reference ID/Investigator# 39818, Tokyo
  - Site Reference ID/Investigator# 39819, Tokyo
  - Site Reference ID/Investigator# 39820, Tokyo
  - Site Reference ID/Investigator# 39821, Tokyo
  - Site Reference ID/Investigator# 39822, Tokyo
  - Site Reference ID/Investigator# 39823, Tokyo
  - Site Reference ID/Investigator# 39824, Tokyo
  - Site Reference ID/Investigator# 39825, Tokyo
  - Site Reference ID/Investigator# 39826, Tokyo
  - Site Reference ID/Investigator# 39827, Tokyo
  - Site Reference ID/Investigator# 39828, Tokyo
  - Site Reference ID/Investigator# 39829, Tokyo
  - Site Reference ID/Investigator# 39830, Tokyo
  - Site Reference ID/Investigator# 39831, Tokyo
  - Site Reference ID/Investigator# 39832, Tokyo
  - Site Reference ID/Investigator# 39833, Tokyo
  - Site Reference ID/Investigator# 39834, Tokyo
  - Site Reference ID/Investigator# 39835, Tokyo
  - Site Reference ID/Investigator# 39836, Tokyo
  - Site Reference ID/Investigator# 39837, Tokyo
  - Site Reference ID/Investigator# 39838, Tokyo
  - Site Reference ID/Investigator# 39894, Tokyo
  - Site Reference ID/Investigator# 39895, Tokyo
  - Site Reference ID/Investigator# 39896, Tokyo
  - Site Reference ID/Investigator# 39897, Tokyo
  - Site Reference ID/Investigator# 39898, Tokyo
  - Site Reference ID/Investigator# 39899, Tokyo
  - Site Reference ID/Investigator# 39900, Tokyo
  - Site Reference ID/Investigator# 39902, Tokyo
  - Site Reference ID/Investigator# 39903, Tokyo
  - Site Reference ID/Investigator# 39904, Tokyo
  - Site Reference ID/Investigator# 39905, Tokyo
  - Site Reference ID/Investigator# 39906, Tokyo
  - Site Reference ID/Investigator# 39907, Tokyo
  - Site Reference ID/Investigator# 39908, Tokyo
  - Site Reference ID/Investigator# 39909, Tokyo
  - Site Reference ID/Investigator# 39911, Tokyo
  - Site Reference ID/Investigator# 39923, Tokyo
  - Site Reference ID/Investigator# 39927, Tokyo
  - Site Reference ID/Investigator# 42718, Tokyo
  - Site Reference ID/Investigator# 42722, Tokyo
  - Site Reference ID/Investigator# 42741, Tokyo
  - Site Reference ID/Investigator# 42742, Tokyo
  - Site Reference ID/Investigator# 42749, Tokyo
  - Site Reference ID/Investigator# 42792, Tokyo
  - Site Reference ID/Investigator# 42795, Tokyo
  - Site Reference ID/Investigator# 42796, Tokyo
  - Site Reference ID/Investigator# 42800, Tokyo
  - Site Reference ID/Investigator# 42860, Tokyo
  - Site Reference ID/Investigator# 42861, Tokyo
  - Site Reference ID/Investigator# 42862, Tokyo
  - Site Reference ID/Investigator# 42863, Tokyo
  - Site Reference ID/Investigator# 42864, Tokyo
  - Site Reference ID/Investigator# 42865, Tokyo
  - Site Reference ID/Investigator# 42891, Tokyo
  - Site Reference ID/Investigator# 58545, Tokyo
  - Site Reference ID/Investigator# 58606, Tokyo
  - Site Reference ID/Investigator# 58610, Tokyo
  - Site Reference ID/Investigator# 58659, Tokyo
  - Site Reference ID/Investigator# 58660, Tokyo
  - Site Reference ID/Investigator# 58661, Tokyo
  - Site Reference ID/Investigator# 58662, Tokyo
  - Site Reference ID/Investigator# 58663, Tokyo
  - Site Reference ID/Investigator# 58664, Tokyo
  - Site Reference ID/Investigator# 58665, Tokyo
  - Site Reference ID/Investigator# 58666, Tokyo
  - Site Reference ID/Investigator# 58667, Tokyo
  - Site Reference ID/Investigator# 58789, Tokyo
  - Site Reference ID/Investigator# 58790, Tokyo
  - Site Reference ID/Investigator# 58798, Tokyo
  - Site Reference ID/Investigator# 58804, Tokyo
  - Site Reference ID/Investigator# 58807, Tokyo
  - Site Reference ID/Investigator# 58809, Tokyo
  - Site Reference ID/Investigator# 58828, Tokyo
  - Site Reference ID/Investigator# 58829, Tokyo
  - Site Reference ID/Investigator# 58830, Tokyo
  - Site Reference ID/Investigator# 36170, Tottori
  - Site Reference ID/Investigator# 36661, Tottori
  - Site Reference ID/Investigator# 36806, Tottori
  - Site Reference ID/Investigator# 36916, Tottori
  - Site Reference ID/Investigator# 39919, Tottori
  - Site Reference ID/Investigator# 39921, Tottori
  - Site Reference ID/Investigator# 39922, Tottori
  - Site Reference ID/Investigator# 39925, Tottori
  - Site Reference ID/Investigator# 39926, Tottori
  - Site Reference ID/Investigator# 42721, Tottori
  - Site Reference ID/Investigator# 36309, Toyama
  - Site Reference ID/Investigator# 36310, Toyama
  - Site Reference ID/Investigator# 36311, Toyama
  - Site Reference ID/Investigator# 36312, Toyama
  - Site Reference ID/Investigator# 36313, Toyama
  - Site Reference ID/Investigator# 36314, Toyama
  - Site Reference ID/Investigator# 36315, Toyama
  - Site Reference ID/Investigator# 36316, Toyama
  - Site Reference ID/Investigator# 36443, Toyama
  - Site Reference ID/Investigator# 36564, Toyama
  - Site Reference ID/Investigator# 36807, Toyama
  - Site Reference ID/Investigator# 36938, Toyama
  - Site Reference ID/Investigator# 39920, Toyama
  - Site Reference ID/Investigator# 39924, Toyama
  - Site Reference ID/Investigator# 39928, Toyama
  - Site Reference ID/Investigator# 39929, Toyama
  - Site Reference ID/Investigator# 39930, Toyama
  - Site Reference ID/Investigator# 39933, Toyama
  - Site Reference ID/Investigator# 39935, Toyama
  - Site Reference ID/Investigator# 42793, Toyama
  - Site Reference ID/Investigator# 42797, Toyama
  - Site Reference ID/Investigator# 42799, Toyama
  - Site Reference ID/Investigator# 42927, Toyama
  - Site Reference ID/Investigator# 58583, Toyama
  - Site Reference ID/Investigator# 58817, Toyama
  - Site Reference ID/Investigator# 58856, Toyama
  - Site Reference ID/Investigator# 58873, Toyama
  - Site Reference ID/Investigator# 36866, Toyohashi
  - Site Reference ID/Investigator# 39308, Tsu
  - Site Reference ID/Investigator# 42713, Tsuyama
  - Site Reference ID/Investigator# 36317, Wakayama
  - Site Reference ID/Investigator# 36318, Wakayama
  - Site Reference ID/Investigator# 36319, Wakayama
  - Site Reference ID/Investigator# 36320, Wakayama
  - Site Reference ID/Investigator# 36321, Wakayama
  - Site Reference ID/Investigator# 36578, Wakayama
  - Site Reference ID/Investigator# 39931, Wakayama
  - Site Reference ID/Investigator# 39932, Wakayama
  - Site Reference ID/Investigator# 39936, Wakayama
  - Site Reference ID/Investigator# 42737, Wakayama
  - Site Reference ID/Investigator# 42906, Wakayama
  - Site Reference ID/Investigator# 58568, Wakayama
  - Site Reference ID/Investigator# 58787, Wakayama
  - Site Reference ID/Investigator# 36592, Yamagata
  - Site Reference ID/Investigator# 36833, Yamagata
  - Site Reference ID/Investigator# 36935, Yamagata
  - Site Reference ID/Investigator# 36952, Yamagata
  - Site Reference ID/Investigator# 39934, Yamagata
  - Site Reference ID/Investigator# 42873, Yamagata
  - Site Reference ID/Investigator# 58599, Yamagata
  - Site Reference ID/Investigator# 58648, Yamagata
  - Site Reference ID/Investigator# 58649, Yamagata
  - Site Reference ID/Investigator# 58650, Yamagata
  - Site Reference ID/Investigator# 58821, Yamagata
  - Site Reference ID/Investigator# 58822, Yamagata
  - Site Reference ID/Investigator# 36322, Yamaguchi
  - Site Reference ID/Investigator# 36323, Yamaguchi
  - Site Reference ID/Investigator# 36324, Yamaguchi
  - Site Reference ID/Investigator# 36325, Yamaguchi
  - Site Reference ID/Investigator# 36583, Yamaguchi
  - Site Reference ID/Investigator# 36595, Yamaguchi
  - Site Reference ID/Investigator# 36662, Yamaguchi
  - Site Reference ID/Investigator# 36797, Yamaguchi
  - Site Reference ID/Investigator# 36904, Yamaguchi
  - Site Reference ID/Investigator# 36917, Yamaguchi
  - Site Reference ID/Investigator# 39937, Yamaguchi
  - Site Reference ID/Investigator# 39938, Yamaguchi
  - Site Reference ID/Investigator# 39939, Yamaguchi
  - Site Reference ID/Investigator# 39940, Yamaguchi
  - Site Reference ID/Investigator# 39941, Yamaguchi
  - Site Reference ID/Investigator# 39942, Yamaguchi
  - Site Reference ID/Investigator# 39943, Yamaguchi
  - Site Reference ID/Investigator# 39944, Yamaguchi
  - Site Reference ID/Investigator# 39945, Yamaguchi
  - Site Reference ID/Investigator# 39947, Yamaguchi
  - Site Reference ID/Investigator# 39949, Yamaguchi
  - Site Reference ID/Investigator# 39950, Yamaguchi
  - Site Reference ID/Investigator# 39952, Yamaguchi
  - Site Reference ID/Investigator# 39953, Yamaguchi
  - Site Reference ID/Investigator# 39954, Yamaguchi
  - Site Reference ID/Investigator# 42732, Yamaguchi
  - Site Reference ID/Investigator# 42735, Yamaguchi
  - Site Reference ID/Investigator# 42794, Yamaguchi
  - Site Reference ID/Investigator# 42842, Yamaguchi
  - Site Reference ID/Investigator# 42843, Yamaguchi
  - Site Reference ID/Investigator# 58578, Yamaguchi
  - Site Reference ID/Investigator# 58714, Yamaguchi
  - Site Reference ID/Investigator# 58808, Yamaguchi
  - Site Reference ID/Investigator# 58863, Yamaguchi
  - Site Reference ID/Investigator# 58864, Yamaguchi
  - Site Reference ID/Investigator# 36695, Yamanashi
  - Site Reference ID/Investigator# 39951, Yamanashi
  - Site Reference ID/Investigator# 39955, Yamanashi
  - Site Reference ID/Investigator# 39956, Yamanashi
  - Site Reference ID/Investigator# 39957, Yamanashi
  - Site Reference ID/Investigator# 39958, Yamanashi
  - Site Reference ID/Investigator# 39959, Yamanashi
  - Site Reference ID/Investigator# 39960, Yamanashi
  - Site Reference ID/Investigator# 39961, Yamanashi
  - Site Reference ID/Investigator# 39962, Yamanashi
  - Site Reference ID/Investigator# 39963, Yamanashi
  - Site Reference ID/Investigator# 58827, Yamanashi
  - Site Reference ID/Investigator# 36239, Yokohama
  - Site Reference ID/Investigator# 39701, Yokohama
  - Site Reference ID/Investigator# 39702, Yokohama
  - Site Reference ID/Investigator# 39703, Yokohama
  - Site Reference ID/Investigator# 39704, Yokohama
  - Site Reference ID/Investigator# 39715, Yokohama
  - Site Reference ID/Investigator# 39357, Yufu
  - Site Reference ID/Investigator# 39358, Yufu

REFERENCES:
- [Derived] Koike T, Harigai M, Ishiguro N, Inokuma S, Takei S, Takeuchi T, Yamanaka H, Takasaki Y, Mimori T, Hiramatsu K, Komatsu S, Tanaka Y. Effect of Methotrexate Plus Adalimumab on the Achievement of Rheumatoid Arthritis Therapeutic Goals: Post Hoc Analysis of Japanese Patients (MELODY Study). Rheumatol Ther. 2016 Jun;3(1):129-141. doi: 10.1007/s40744-015-0023-x. Epub 2015 Dec 22. PMID 27747511
- [Derived] Koike T, Harigai M, Ishiguro N, Inokuma S, Takei S, Takeuchi T, Yamanaka H, Haruna S, Ushida N, Kawana K, Tanaka Y. Safety and effectiveness of adalimumab in Japanese rheumatoid arthritis patients: postmarketing surveillance report of 7740 patients. Mod Rheumatol. 2014 May;24(3):390-8. doi: 10.3109/14397595.2013.843760. Epub 2013 Nov 6. PMID 24252049

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The sponsor was required to include all patients diagnosed with rheumatoid arthritis and who were treated Humira in routine medical practice during the review period by the Pharmaceuticals and Medical Devices Agency (PMDA).
Pre-assignment Details: The study was completed when the PMDA had completed their review. A total of 7972 patients were registered and case report forms were retrieved for 7891 patients; 151 patients were excluded from the analysis because the case report forms were either duplicated (n=150) or the patient was included in another survey (n=1).
Groups:
- Humira: Patients who received Humira for 24 weeks during the PMDA review period.
Period: Overall Study
Arm/Group | Humira
Started | 7740
Completed | 5490
Not Completed | 2250
Not completed — Adverse Event | 767
Not completed — Lack of Efficacy | 849
Not completed — Non-compliance | 274
Not completed — Lost to Follow-up | 241
Not completed — Other | 119

BASELINE CHARACTERISTICS:
Arm/Group | Humira
Number analyzed (Participants) | 7740
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (13.0)
Age, Customized [Number; unit: participants]
  <20 years | 26
  >=20-<30 | 165
  >=30-<40 | 461
  >=40-<50 | 828
  >=50-<60 | 1803
  >=60-<70 | 2515
  >=70-<80 | 1676
  >=80-<90 | 261
  >=90 | 4
  No data | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6388
  Male | 1352
Region of Enrollment [Number; unit: participants]
  Japan | 7740

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Patients With Adverse Events
Description: Adverse events were assessed from the time treatment began until treatment ended after 24 weeks. Details about the adverse events and serious adverse events are presented with the adverse event section of the disclosure. This outcome is measured as a percentage of patients with adverse events.
Time Frame: Baseline to Week 24
Population: The safety population included all patients who received at least one dose of Humira, had one set of case report forms, and were registered with PMDA during the review period.
Measure: Number; unit: Percentage of Patients
Arm/Group | Humira
Number analyzed (Participants) | 7740
Percentage of Patients | 27.8

2. Secondary Outcome: Physicians' Overall Effectiveness Response Rating
Description: Physicians' rated the level of overall patient improvement as "markedly improved," "improved," "not changed," or "not assessable" by comparing clinical conditions at Week 24 or at discontinuation with baseline conditions.
Time Frame: Week 24
Population: Of the 7740 subjects treated, 938 patients were removed; 16 patients used Humira for another indication label, 812 patients had data missing at baseline or at least 1 other time point, and 254 patients were treated with Humira for less than 2 weeks. Patients may have been in more than 1 category.
Measure: Number; unit: Percentage of Patients
Groups:
- Physician Response Rating: The full analysis set was used to determine the physicians' overall response rating.
Arm/Group | Physician Response Rating
Number analyzed (Participants) | 6802
Percentage of Patients
  Markedly Improved | 29.1
  Improved | 45.2
  Not Changed | 19.6
  Not Assessable | 6.1

3. Primary Outcome: Patient Effectiveness Response Rating and Effective Rate of Humira With Disease Activity Score (DAS) 28 at Week 4
Description: Effectiveness was assessed according to European League Against Rheumatism (EULAR) response criteria. The investigator rated patient response as good, moderate, or none from baseline to Week 4. The DAS 28 index is a measure of activity derived from the number of swollen or tender joints, laboratory tests of inflammation, and patient assessment of global health (10 cm line ranging from very good to very bad).
Time Frame: Week 4
Population: Of the 7740 subjects treated, 938 patients were removed; 16 patients used Humira for another indication, 812 patients had data missing at baseline or at least 1 other time point, and 254 patients were treated with Humira for less than 2 weeks. Patients may have been in more than 1 category.
Measure: Number; unit: Percentage of patients
Groups:
- Humira - Good Response: Patients who received Humira during the PMDA review period and had a good response according to DAS 28 (improvement > 1.2) at Week 4. All variables may not have been tested; therefore, a patient may not have been included.
- Humira - Moderate Response: Patients who received Humira during the PMDA review period and had a moderate response according to DAS 28 (improvement 0.6 to 1.2) at Week 4. All variables may not have been tested; therefore, a patient may not have been included.
- Humira - No Response: Patients who received Humira during the PMDA review period and had no response according to DAS 28 (improvement <0.6) at Week 4. All variables may not have been tested; therefore, a patient may not have been included.
- Effective Rate-Sum of Patients With Good or Moderate Response: Patients who received Humira during the PMDA review period and had a moderate or good response to DAS 28 (improvement =>0.6) at Week 4. All variables may not have been tested; therefore, a patient may not have been included.
Arm/Group | Humira - Good Response | Humira - Moderate Response | Humira - No Response | Effective Rate-Sum of Patients With Good or Moderate Response
Number analyzed (Participants) | 3341 | 3341 | 3341 | 3341
Percentage of patients | 20.4 | 45.7 | 33.9 | 66.1

4. Primary Outcome: Patient Effectiveness Response Rating and Effective Rate of Humira With DAS 28 at Week 12
Description: Effectiveness was assessed according to European League Against Rheumatism (EULAR) response criteria. The investigator rated patient response as good, moderate, or none from baseline to Week 12. The DAS 28 index is a measure of activity derived from the number of swollen or tender joints, laboratory tests of inflammation, and patient assessment of global health (10 cm line ranging from very good to very bad).
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: percentage of patients
Groups:
- Humira - Good Response: Patients who received Humira during the PMDA review period and had a good response to DAS 28 (improvement > 1.2) at Week 12. All variables may not have been tested; therefore, a patient may not have been included.
- Humira - Moderate Response: Patients who received Humira during the PMDA review period and had a moderate response to DAS 28 (improvement 0.6 to 1.2) at Week 12. All variables may not have been tested; therefore, a patient may not have been included.
- Humira - No Response: Patients who received Humira during the PMDA review period and had no response to DAS 28 (improvement < 0.6) at Week 12. All variables may not have been tested; therefore, a patient may not have been included.
- Effective Rate-Sum of Patients With Good or Moderate Response: Patients who received Humira during the PMDA review period and had a moderate or good response to DAS 28 (improvement =>0.6) at Week 12. All variables may not have been tested; therefore, a patient may not have been included.
Arm/Group | Humira - Good Response | Humira - Moderate Response | Humira - No Response | Effective Rate-Sum of Patients With Good or Moderate Response
Number analyzed (Participants) | 3927 | 3927 | 3927 | 3927
percentage of patients | 26.4 | 42.6 | 31.1 | 68.9

5. Primary Outcome: Patient Effectiveness Response Rating and Effective Rate of Humira With DAS 28 at Week 24
Description: Effectiveness was assessed according to European League Against Rheumatism (EULAR) response criteria. The investigator rated patient response as good, moderate, or none from baseline to Week 24. The DAS 28 index is a measure of activity derived from the number of swollen or tender joints, laboratory tests of inflammation, and patient assessment of global health (10 cm line ranging from very good to very bad).
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: Percentage of Patients
Groups:
- Humira - Good Response: Patients who received Humira during the PMDA review period and had a good response to DAS 28 (improvement > 1.2) at Week 4.at Week 24. All variables may not have been tested; therefore, a patient may not have been included.
- Humira - Moderate Response: Patients who received Humira during the PMDA review period and had a moderate response to DAS 28 (improvement 0.6 to 1.2) at Week 24. All variables may not have been tested; therefore, a patient may not have been included.
- Humira - No Response: Patients who received Humira during the PMDA review period and had no response to DAS 28 (improvement < 0.6) at Week 24. All variables may not have been tested; therefore, a patient may not have been included.
- Effective Rate-Sum of Patients With Good and Moderate Response: Patients who received Humira during the PMDA review period and had a moderate or good response to DAS 28 (improvement =>0.6) at Week 24. All variables may not have been tested; therefore, a patient may not have been included.
Arm/Group | Humira - Good Response | Humira - Moderate Response | Humira - No Response | Effective Rate-Sum of Patients With Good and Moderate Response
Number analyzed (Participants) | 4410 | 4410 | 4410 | 4410
Percentage of Patients | 30.7 | 39.3 | 29.9 | 70.1

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the time treatment began until treatment ended after 24 weeks.
Arm/Group | Humira
Serious Adverse Events (participants affected / at risk) | 469/7740
Other Adverse Events (participants affected / at risk) | 863/7740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=7740)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 4
Anemia folate deficiency (Blood and lymphatic system disorders) | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3
Lymphadenitis (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Bone Marrow Failure (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 5
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 2
Atrial tachycardia (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 5
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Right ventricular failure (Cardiac disorders) | 1
Sick sinus syndrome (Cardiac disorders) | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Retinal vein occlusion (Eye disorders) | 1
Scleritis (Eye disorders) | 1
Uveitis (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Colitis ischemic (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Gastric ulcer hemorrhage (Gastrointestinal disorders) | 2
Gastric ulcer perforation (Gastrointestinal disorders) | 1
Gastritis atrophic (Gastrointestinal disorders) | 1
Gastritis hemorrhagic (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal necrosis (Gastrointestinal disorders) | 1
Ileitis (Gastrointestinal disorders) | 1
Ileus paralytic (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Melena (Gastrointestinal disorders) | 2
Esophageal ulcer (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 2
Peritonitis (Gastrointestinal disorders) | 1
Small intestine ulcer (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Duodenal stenosis (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Diverticular perforation (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 3
Death (General disorders) | 4
Device breakage (General disorders) | 1
Drowning (General disorders) | 1
Gait disturbance (General disorders) | 1
Hyperthermia (General disorders) | 1
Local swelling (General disorders) | 1
Malaise (General disorders) | 2
Multiorgan failure (General disorders) | 2
Edema (General disorders) | 1
Edema peripheral (General disorders) | 1
Pyrexia (General disorders) | 13
Cholecystitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Hepatic failure (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 4
Hepatitis (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Liver disorder (Hepatobiliary disorders) | 2
Gallbladder polyp (Hepatobiliary disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Anaphylactoid reaction (Immune system disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Bronchiolitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Bronchopneumonia (Infections and infestations) | 5
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 12
Cystitis (Infections and infestations) | 2
Disseminated tuberculosis (Infections and infestations) | 1
Endophthalmitis (Infections and infestations) | 1
Erysipelas (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 4
Hepatitis B (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 12
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Lymph node tuberculosis (Infections and infestations) | 1
Meningitis (Infections and infestations) | 1
Meningitis aseptic (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 1
Peritonsillar abscess (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 41
Pneumonia chlamydial (Infections and infestations) | 2
Pneumonia cytomegaloviral (Infections and infestations) | 2
Pneumonia legionella (Infections and infestations) | 3
Pneumonia pneumococcal (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 1
Pseudomembranous colitis (Infections and infestations) | 1
Pulmonary tuberculosis (Infections and infestations) | 3
Pulpitis dental (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 4
Pyelonephritis acute (Infections and infestations) | 1
Pyothorax (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 2
Sepsis (Infections and infestations) | 13
Septic shock (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Tuberculous pleurisy (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 4
Muscle abscess (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 2
Arthritis bacterial (Infections and infestations) | 7
Peritoneal tuberculosis (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Wound abscess (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 13
Bursitis infective (Infections and infestations) | 2
Lung infection (Infections and infestations) | 1
Tuberculosis gastrointestinal (Infections and infestations) | 1
Atypical mycobacterial infection (Infections and infestations) | 1
Enterocolitis viral (Infections and infestations) | 1
Purulence (Infections and infestations) | 1
Mycobacterial infection (Infections and infestations) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 26
Device related infection (Infections and infestations) | 1
Enterocolitis bacterial (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Pneumonia cryptococcal (Infections and infestations) | 2
Compression fracture (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 10
Femur fracture (Injury, poisoning and procedural complications) | 5
Fibula fracture (Injury, poisoning and procedural complications) | 2
Foot fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 6
Subdural hematoma (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 6
Tibia fracture (Injury, poisoning and procedural complications) | 1
Ulna fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Joint injury (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 3
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood glucose increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
C-reactive protein increased (Investigations) | 2
Carcinoembryonic antigen increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Blood beta-D-glucan abnormal (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Cell marker increased (Investigations) | 1
Candida test positive (Investigations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypoglycemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatic (Musculoskeletal and connective tissue disorders) | 1
Polymyositis (Musculoskeletal and connective tissue disorders) | 3
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2
Foot deformity (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung squamous cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Gallbladder cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Cauda equina syndrome (Nervous system disorders) | 1
Cerebellar infarction (Nervous system disorders) | 1
Cerebral hemorrhage (Nervous system disorders) | 3
Cerebral thrombosis (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 1
Demyelination (Nervous system disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Subarachnoid hemorrhage (Nervous system disorders) | 5
Syncope (Nervous system disorders) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Putamen hemorrhage (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Cerebral infarction (Nervous system disorders) | 4
Completed suicide (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 1
Calculus ureteric (Renal and urinary disorders) | 1
Nephrotic syndrome (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 3
Renal impairment (Renal and urinary disorders) | 2
Henoch-Schonlein purpura nephritis (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 40
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1
Diffuse panbronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Rash erythematosus (Skin and subcutaneous tissue disorders) | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Generalized erythema (Skin and subcutaneous tissue disorders) | 1
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 1
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral circulatory failure (Vascular disorders) | 1
Shock (Vascular disorders) | 1
Vasculitis (Vascular disorders) | 1
Vasculitis necrotizing (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Arterial hemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Humira (N=7740)
Injection site erythema (General disorders) | 160
Injection site reaction (General disorders) | 108
Pyrexia (General disorders) | 99
Hepatic function abnormal (Hepatobiliary disorders) | 110
Nasopharyngitis (Infections and infestations) | 94
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 79
Pruritus (Skin and subcutaneous tissue disorders) | 78
Rash (Skin and subcutaneous tissue disorders) | 255

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.